CLINICAL TRIAL: NCT03970837
Title: A 52-week, Phase 3, Multicentre, Randomised, Double Blind, Efficacy and Safety Study, Comparing GSK3196165 With Placebo and With Tofacitinib in Combination With Conventional Synthetic DMARDs, in Participants With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Conventional Synthetic DMARDs or Biologic DMARDs
Brief Title: Efficacy and Safety of GSK3196165 Versus Placebo and Tofacitinib in Participants With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Conventional Synthetic (cs)/Biologic (b) Disease Modifying Anti-rheumatic Drugs (DMARDs)
Acronym: contRAst 2
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Only Asia cohort is early terminated.Limited efficacy demonstrated in the contRAst program does not support a suitable benefit/risk profile for otilimab as a potential treatment for RA. GSK has decided not to progress with regulatory submissions.
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201791
Record Dates: First submitted 2019-05-16; First posted 2019-06-03 (Actual); Results first posted 2023-11-30 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; GSK3196165; Otilimab; Tofacitinib; Placebo; DMARDs
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Otilimab; tofacitinib

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of six intervention arms in ratio of 6:6:3:1:1:1
Who Masked: Participant, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- GSK3196165 90mg + csDMARD (Global Cohort) (Experimental): Participants in Global Cohort received GSK3196165 90 mg subcutaneous (SC) injection once weekly for 52 weeks in combination with conventional synthetic disease-modifying antirheumatic drugs (csDMARD).
  Interventions: Biological: GSK3196165 (Otilimab)
- GSK3196165 150mg + csDMARD (Global Cohort) (Experimental): Participants in Global Cohort received GSK3196165 150 mg subcutaneous (SC) injection once weekly for 52 weeks in combination with csDMARD.
  Interventions: Biological: GSK3196165 (Otilimab)
- Tofacitinib 5mg + csDMARD (Global Cohort) (Active Comparator): Participants in Global Cohort received Tofacitinib 5mg capsule, orally, twice daily (BID) in combination with csDMARD plus placebo injection weekly to maintain the blind for 52 weeks.
  Interventions: Drug: Tofacitinib
- Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) (Placebo Comparator): Participants in Global Cohort received Placebo weekly SC injection in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo to GSK3196165 90 mg, SC injection, once weekly in combination with csDMARD until 52 weeks.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo
- Placebo +csDMARD and GSK3196165 150mg +csDMARD (Global Cohort) (Placebo Comparator): Participants in Global Cohort received Placebo weekly SC injection in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo to GSK3196165 150 mg, SC injection, once weekly in combination with csDMARD until 52 weeks.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo
- Placebo +csDMARD and Tofacitinib 5mg +csDMARD (Global Cohort) (Placebo Comparator): Participants in Global Cohort received Placebo capsule BID in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo capsule to Tofacitinib 5mg, capsule, orally, BID in combination with csDMARD plus placebo injection to maintain the blind for 52 weeks.
  Interventions: Drug: Tofacitinib; Drug: Placebo
- GSK3196165 90mg + csDMARD (Asia Cohort) (Experimental): Participants in Asia Cohort received GSK3196165 90 mg subcutaneous (SC) injection once weekly for 52 weeks in combination with csDMARD.
  Interventions: Biological: GSK3196165 (Otilimab)
- GSK3196165 150mg + csDMARD (Asia Cohort) (Experimental): Participants in Asia Cohort received GSK3196165 150 mg subcutaneous (SC) injection once weekly for 52 weeks in combination with csDMARD.
  Interventions: Biological: GSK3196165 (Otilimab)
- Tofacitinib 5mg + csDMARD (Asia Cohort) (Active Comparator): Participants in Asia Cohort received Tofacitinib 5mg capsule, orally, twice daily (BID) in combination with csDMARD plus placebo injection weekly to maintain the blind for 52 weeks.
  Interventions: Drug: Tofacitinib
- Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) (Placebo Comparator): Participants in Asia Cohort received Placebo weekly SC injection in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo to GSK3196165 90 mg, SC injection, once weekly in combination with csDMARD until 52 weeks.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo
- Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) (Placebo Comparator): Participants in Asia Cohort received Placebo weekly SC injection in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo to GSK3196165 150 mg, SC injection, once weekly in combination with csDMARD until 52 weeks.
  Interventions: Biological: GSK3196165 (Otilimab); Drug: Placebo
- Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort) (Placebo Comparator): Participants in Asia Cohort received Placebo capsule BID in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo capsule to Tofacitinib 5mg, capsule, orally, BID in combination with csDMARD plus placebo injection to maintain the blind for 52 weeks.
  Interventions: Drug: Tofacitinib; Drug: Placebo

INTERVENTIONS:
Biological: GSK3196165 (Otilimab) — GSK3196165 solution in vial/pre-filled syringe (PFS) was administered SC.
  Arms: GSK3196165 150mg + csDMARD (Asia Cohort); GSK3196165 150mg + csDMARD (Global Cohort); GSK3196165 90mg + csDMARD (Asia Cohort); GSK3196165 90mg + csDMARD (Global Cohort); Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort); Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort); Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort); Placebo +csDMARD and GSK3196165 150mg +csDMARD (Global Cohort)
Drug: Tofacitinib — Tofacitinib capsule (over encapsulated 5mg tablet) was administered orally.
  Arms: Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort); Placebo +csDMARD and Tofacitinib 5mg +csDMARD (Global Cohort); Tofacitinib 5mg + csDMARD (Asia Cohort); Tofacitinib 5mg + csDMARD (Global Cohort)
Drug: Placebo — Placebo matching GSK3196165 and Tofacitinib was administered.
  Arms: Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort); Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort); Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort); Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort); Placebo +csDMARD and GSK3196165 150mg +csDMARD (Global Cohort); Placebo +csDMARD and Tofacitinib 5mg +csDMARD (Global Cohort)

SUMMARY:
This study [contRAst 2 (201791: NCT03970837)] is a phase 3, randomized, multicenter, double blind study to assess the safety and efficacy of GSK3196165 in combination with csDMARD(s), for the treatment of adult participants with moderate to severe active rheumatoid arthritis (RA) who have had an inadequate response to csDMARD(s) or bDMARD(s). The study will consist of a screening phase of up to 6 weeks followed by a 52 week treatment phase in which participants will be randomized in a ratio of 6:6:3:1:1:1 to receive GSK3196165 150 milligrams (mg) subcutaneous (SC) weekly, GSK3196165 90 mg SC weekly, tofacitinib capsules (cap) 5 mg twice a day or placebo (three arms, each placebo arm will have 12 weeks placebo followed by 40 weeks active treatment) respectively, all in combination with csDMARD(s). Participants who, in investigator's judgement will benefit from extended treatment with GSK3196165 may be included in the long-term extension study [contRAst X (209564: NCT04333147)]. For those participants who do not continue into the long term-extension study, there will be an 8 week safety follow-up visit following the treatment phase.

ELIGIBILITY:
Key inclusion criteria

* >=18 years of age
* Has had RA for >=6 months and was not diagnosed before 16 years of age
* Has active disease, as defined by having both*

  * >=6/68 tender/painful joint count (TJC), and
  * >=6/66 swollen joint count (SJC)
* Has at least 1 bone erosion present on hand/wrist or foot radiographs
* Has had an inadequate response to one or two of the csDMARDs:

  * methotrexate (MTX) 15-25 mg/week** oral or injected
  * hydroxychloroquine up to 400 mg/day or chloroquine up to 250 mg/day
  * sulfasalazine up to 3000 mg/day
  * leflunomide up to 20 mg/day***
  * bucillamine up to 100 mg/day (or up to 300 mg/day if permitted per local requirement)
  * iguratimod up to 50 mg/day

    * If surgical treatment of a joint has been performed, that joint cannot be counted in the TJC or SJC.

      * A lower dose of 7.5 mg/week is acceptable if reduced for reasons of intolerance to MTX or per local requirement.

        * Concomitant use of leflunomide and methotrexate is not allowed, for safety reasons.

Key exclusion criteria

* History of other inflammatory rheumatologic or systemic autoimmune disorder, other than Sjögren's syndrome secondary to RA, that may confound the evaluation of the effect of the study intervention.
* Has had any active and/or recurrent infections (excluding recurrent fungal infections of the nail bed) or has required management of acute or chronic infections.
* Has received prior treatment with an antagonist of GM-CSF or its receptor or Janus kinase (JAK) inhibitors (either experimental or approved).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1764 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (202):
- United States (61):
  - GSK Investigational Site, Flagstaff, Arizona
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Poway, California
  - GSK Investigational Site, Riverside, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, Tustin, California
  - GSK Investigational Site, Van Nuys, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Collins, Colorado
  - GSK Investigational Site, Aventura, Florida
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Daytona Beach, Florida
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Margate, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, New Port Richey, Florida
  - GSK Investigational Site, Palmetto Bay, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tamarac, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Idaho Falls, Idaho
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bowling Green, Kentucky
  - GSK Investigational Site, Lake Charles, Louisiana
  - GSK Investigational Site, Monroe, Louisiana
  - GSK Investigational Site, Hagerstown, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Grand Blanc, Michigan
  - GSK Investigational Site, Lansing, Michigan
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, Freehold, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Brooklyn, New York
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Minot, North Dakota
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Yukon, Oklahoma
  - GSK Investigational Site, Duncansville, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Wyomissing, Pennsylvania
  - GSK Investigational Site, Columbia, South Carolina
  - GSK Investigational Site, Myrtle Beach, South Carolina
  - GSK Investigational Site, Summerville, South Carolina
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Amarillo, Texas
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Colleyville, Texas
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Lubbock, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Tomball, Texas
  - GSK Investigational Site, Glendale, Wisconsin
- Argentina (8):
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, San Miguel de Tucumán, Tucumán Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma Buenos Aires
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, San Juan
- Australia (6):
  - GSK Investigational Site, Westmead, New South Wales
  - GSK Investigational Site, Gold Coast, Queensland
  - GSK Investigational Site, Woodville, South Australia
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Box Hill, Victoria
  - GSK Investigational Site, Heidelberg West, Victoria
- Bulgaria (8):
  - GSK Investigational Site, Blagoevgrad
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Rousse
  - GSK Investigational Site, Sevlievo
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Stara Zagora
  - GSK Investigational Site, Vidin
- China (29):
  - GSK Investigational Site, Bengbu, Anhui
  - GSK Investigational Site, Guilin, Guangxi
  - GSK Investigational Site, Shijiazhuang, Hebei
  - GSK Investigational Site, Wuhan, Hubei
  - GSK Investigational Site, Changsha, Hunan
  - GSK Investigational Site, Zhuzhou, Hunan
  - GSK Investigational Site, Baotou, Inner Mongolia
  - GSK Investigational Site, Tongliao, Inner Mongolia
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Taizhou, Jiangsu
  - GSK Investigational Site, Xuzhou, Jiangsu
  - GSK Investigational Site, Yancheng, Jiangsu
  - GSK Investigational Site, Jiujiang, Jiangxi
  - GSK Investigational Site, Nanchang, Jiangxi
  - GSK Investigational Site, Changchun, Jilin
  - GSK Investigational Site, Jinzhou, Liaoning
  - GSK Investigational Site, Huzhou, Zhejiang
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Changchun
  - GSK Investigational Site, Changzhou
  - GSK Investigational Site, Chengdu
  - GSK Investigational Site, Guangzhou
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Nanjing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin
  - GSK Investigational Site, Xi'an
  - GSK Investigational Site, Yangzhou
  - GSK Investigational Site, Yanji
- Colombia (4):
  - GSK Investigational Site, Barranquilla
  - GSK Investigational Site, Bogotá
  - GSK Investigational Site, Bucaramanga
  - GSK Investigational Site, Medellín
- Estonia (3):
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- GSK Investigational Site, Cahors, France
- Germany (5):
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Rendsburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Magdeburg
- Hungary (3):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Szentes
  - GSK Investigational Site, Székesfehérvár
- Japan (24):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Hyōgo
  - GSK Investigational Site, Ibaraki
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kagoshima
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Kochi
  - GSK Investigational Site, Kumamoto
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagano
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Niigata
  - GSK Investigational Site, Okayama
  - GSK Investigational Site, Saga
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Shizuoka
  - GSK Investigational Site, Tokyo
  - GSK Investigational Site, Tottori
  - GSK Investigational Site, Wakayama
  - GSK Investigational Site, Yamaguchi
- Mexico (4):
  - GSK Investigational Site, Mexico City, Durango
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Mérida, Yucatán
  - GSK Investigational Site, San Luis Potosí City
- Poland (18):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bydgoszcz
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Grodzisk Mazowiecki
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Nowy Targ
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Poznan
  - GSK Investigational Site, Siedlce
  - GSK Investigational Site, Sochaczew
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (11):
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Korolyov
  - GSK Investigational Site, Krasnoyarsk
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ulyanovsk
  - GSK Investigational Site, Yaroslavl
  - GSK Investigational Site, Yekaterinburg
- South Korea (8):
  - GSK Investigational Site, Anyang-Si, Gyeonggi-do
  - GSK Investigational Site, Cheonan-si
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seongnam-si
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Santander
  - GSK Investigational Site, Seville
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Muang
  - GSK Investigational Site, Rajathevee
- United Kingdom (3):
  - GSK Investigational Site, Romford, Essex
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Kenilworth, Warwickshire

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Fleischmann RM, van der Heijde D, Strand V, Atsumi T, McInnes IB, Takeuchi T, Taylor PC, Bracher M, Brooks D, Davies J, Goode C, Gupta A, Mukherjee S, O'Shea C, Saurigny D, Schifano LA, Shelton C, Smith JE, Wang M, Wang R, Watts S, Weinblatt ME. Anti-GM-CSF otilimab versus tofacitinib or placebo in patients with active rheumatoid arthritis and an inadequate response to conventional or biologic DMARDs: two phase 3 randomised trials (contRAst 1 and contRAst 2). Ann Rheum Dis. 2023 Dec;82(12):1516-1526. doi: 10.1136/ard-2023-224482. Epub 2023 Sep 12. PMID 37699654
- See also: 209564 contRAst X NCT04333147 — https://clinicaltrials.gov/ct2/show/NCT04333147?term=209564&draw=2&rank=1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: For both Global and Asia cohorts, participants were randomized in a ratio of 6:6:3:1:1:1 to GSK3196165 90 milligram (mg):GSK3196165 150mg:Tofacitinib 5mg:Placebo:Placebo:Placebo. At Week 12, participants randomized to three placebo arms switched to active intervention arms (GSK3196165 90mg, 150mg or Tofacitinib 5mg), receiving the active intervention for 40 weeks. Participants who were randomized to active intervention arms from study day 1, received the active intervention for 52 weeks.
Pre-assignment Details: Total of 1764 participants were enrolled in the study (1625 in Global and 139 in Asia cohorts which is supplementary to Global Cohort). One participant from GSK3196165 150mg (Asia cohort) arm was randomized but not treated. The study was terminated early only for Asia Cohort as the limited efficacy did not support the benefit risk profile of Otilimab as a potential treatment.
Groups:
- Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort): Participants in Global Cohort received Placebo weekly SC injection in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo to GSK3196165 150 mg, SC injection, once weekly in combination with csDMARD until 52 weeks
- Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort): Participants in Global Cohort received Placebo capsule BID in combination with csDMARD for 12 weeks. At week 12, participants were switched from placebo capsule to Tofacitinib 5mg, capsule, orally, BID in combination with csDMARD plus placebo injection to maintain the blind for 52 weeks.
Period: Overall Study
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort) | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Started (All randomized participants who received at least one dose of study treatment. This population will be based on the treatment the participant was randomized to.) | 545 | 539 | 271 | 91 | 89 | 90 | 47 | 49 | 19 | 6 | 8 | 9
Safety Set (All randomized participants who received at least one dose of study treatment. This population will be based on the treatment the participants actually received.) | 545 | 539 | 286 | 0 | 0 | 0 | 47 | 49 | 19 | 0 | 0 | 0
Safety Set-Placebo Switch (All participants randomized to a placebo switch treatment arm (i.e. Placebo to GSK3196165 90mg, Placebo to GSK3196165 150mg or Placebo to Tofacitinib 5mg) who received at least one dose of study treatment after Week 12.) | 0 | 0 | 0 | 85 | 80 | 67 | 0 | 0 | 0 | 6 | 8 | 8
Completed | 461 | 447 | 231 | 73 | 69 | 68 | 25 | 23 | 15 | 4 | 5 | 4
Not Completed | 84 | 92 | 40 | 18 | 20 | 22 | 22 | 26 | 4 | 2 | 3 | 5
Not completed — Adverse Event | 23 | 20 | 16 | 6 | 4 | 5 | 1 | 5 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 14 | 12 | 1 | 2 | 3 | 4 | 6 | 1 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 6 | 5 | 5 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 5 | 8 | 4 | 1 | 5 | 2 | 4 | 5 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 32 | 35 | 12 | 8 | 6 | 8 | 2 | 3 | 0 | 0 | 0 | 1
Not completed — PROTOCOL-SPECIFIED WITHDRAWAL CRITERION MET | 3 | 12 | 2 | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — STUDY TERMINATED BY SPONSOR | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 11 | 2 | 1 | 2 | 3

BASELINE CHARACTERISTICS:
Population: Intent-To-Treat (ITT) Population (All randomized participants who received at least 1 dose of study treatment) was used for Global cohort and ITT-Supplementary Asia Cohort (Participants randomized on or after 07-August-2021 who received at least one dose of study treatment) was used for Asia cohort. One participant from the GSK3196165 150mg + csDMARD (Asia Cohort) arm was randomized but not treated so is excluded from the ITT-Asia cohort population.
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort) | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort) | Total
Number analyzed (Participants) | 545 | 539 | 271 | 91 | 89 | 90 | 47 | 49 | 19 | 6 | 8 | 9 | 1763
Age, Customized [Count of Participants; unit: Participants]
  18-49 Years | 172 | 150 | 79 | 30 | 23 | 23 | 19 | 21 | 3 | 2 | 3 | 3 | 528
  50-64 Years | 254 | 264 | 125 | 47 | 43 | 45 | 23 | 22 | 11 | 3 | 5 | 5 | 847
  >=65 Years | 119 | 125 | 67 | 14 | 23 | 22 | 5 | 6 | 5 | 1 | 0 | 1 | 388
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 431 | 430 | 229 | 68 | 73 | 73 | 34 | 37 | 12 | 4 | 5 | 7 | 1403
  Male | 114 | 109 | 42 | 23 | 16 | 17 | 13 | 12 | 7 | 2 | 3 | 2 | 360
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 29 | 39 | 21 | 6 | 4 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 105
  ASIAN | 96 | 98 | 49 | 16 | 16 | 16 | 47 | 49 | 19 | 6 | 8 | 9 | 429
  BLACK OR AFRICAN AMERICAN | 10 | 8 | 3 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 24
  WHITE | 409 | 393 | 197 | 67 | 69 | 67 | 0 | 0 | 0 | 0 | 0 | 0 | 1202
  MULTIPLE | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  MISSING | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage (%) of Participants With 20% Improvement in American College of Rheumatology Criteria (ACR20) at Week 12 Superiority Comparison With Placebo (Global Cohort)
Description: ACR20 is calculated as a 20% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) [visual analogue scale (VAS) with values from 0=best to 100=worst], Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant [high sensitivity C-reactive Protein milligram per liter (mg/L) (hsCRP)]. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the Intent-to-Treat (ITT) set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Groups:
- Pooled Placebo (Global Cohort): Participants received Placebo weekly SC injection in combination with csDMARD until Week 12. The placebo arms are pooled into a single placebo arm.
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 54.9 | 54.5 | 71.1 | 32.5
Statistical Analysis 1: Comparison: GSK3196165 90mg + csDMARD (Global Cohort) vs Pooled Placebo (Global Cohort); The null hypothesis is defined as there is no difference between the 90mg dose of GSK3196165 and placebo in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 90mg dose of GSK3196165 differs from placebo in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p < 0.0001, Regression, Logistic; OR and corresponding 95% CI for OR are generated from the logistic regression model adjusted for Baseline TJC68, Baseline SJC66 and Treatment Group; Odds Ratio (OR) = 2.57, 95% CI 2-sided [1.87 to 3.53]
Statistical Analysis 2: Comparison: GSK3196165 150mg + csDMARD (Global Cohort) vs Pooled Placebo (Global Cohort); The null hypothesis is defined as there is no difference between the 150mg dose of GSK3196165 and placebo in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 150mg dose of GSK3196165 differs from placebo in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 2.55, 95% CI 2-sided [1.85 to 3.50]
Statistical Analysis 3: Comparison: Tofacitinib 5mg + csDMARD (Global Cohort) vs Pooled Placebo (Global Cohort); The null hypothesis is defined as there is no difference between the 05mg dose of Tofacitinib and placebo in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 05mg dose of Tofacitinib differs from placebo in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 5.38, 95% CI 2-sided [3.66 to 7.90]
Statistical Analysis 4: Comparison: GSK3196165 90mg + csDMARD (Global Cohort) vs Tofacitinib 5mg + csDMARD (Global Cohort); The null hypothesis is defined as there is no difference between the 90 mg dose of GSK3196165 and 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 90 mg dose of GSK3196165 differs from 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.48, 95% CI 2-sided [0.34 to 0.66]
Statistical Analysis 5: Comparison: GSK3196165 150mg + csDMARD (Global Cohort) vs Tofacitinib 5mg + csDMARD (Global Cohort); The null hypothesis is defined as there is no difference between the 150mg dose of GSK3196165 and 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12, versus the alternative hypothesis that the 150mg dose of GSK3196165 differs from 05mg dose of Tofacitinib in the proportion of participants achieving ACR20 response at Week 12; Test type: Superiority; p < 0.0001, Regression, Logistic; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.47, 95% CI 2-sided [0.34 to 0.66]

2. Primary Outcome: Percentage (%) of Participants With 20% Improvement in American College of Rheumatology Criteria (ACR20) at Week 12 (Asia Cohort)
Description: ACR20 is calculated as a 20% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) [visual analogue scale (VAS) with values from 0=best to 100=worst], Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant [high sensitivity C-reactive Protein milligram per liter (mg/L) (hsCRP)]. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: ITT-Supplementary Asia Cohort Population consisted of participants randomized on or after 07-August-2021 who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Number; unit: Percentage of participants
Groups:
- Pooled Placebo (Asia Cohort): Participants in Asia Cohort received Placebo weekly SC injection in combination with csDMARD until Week 12. The placebo arms are pooled into a single placebo arm.
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 44 | 42 | 19 | 21
Percentage of participants | 45.0 | 40.0 | 68.0 | 14.0

3. Secondary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Total Score Less Than or Equal to (<=)10 [CDAI Low Disease Activity (LDA)] at Week 12 (Global Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the ITT set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 26.5 | 25.1 | 36.8 | 11.4

4. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 (Global Cohort)
Description: HAQ-DI is a 20-question instrument that assesses the degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Scores on a scale | -0.32 (0.029) | -0.31 (0.029) | -0.46 (0.037) | -0.14 (0.038)

5. Secondary Outcome: Percentage of Participants Achieving 20% Improvement in ACR20 at Week 24: Non-inferiority Comparison With Tofacitinib (Global Cohort)
Description: ACR20 is calculated as a 20% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) [visual analogue scale (VAS) with values from 0=best to 100=worst], Physician Global Assessment of Arthritis Disease Activity (PhGA) (VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant [high sensitivity C-reactive Protein milligram per liter (mg/L) (hsCRP)].
Time Frame: Week 24
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 52. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants | 65.0 | 62.5 | 79.8
Statistical Analysis 1: Comparison: GSK3196165 90mg + csDMARD (Global Cohort) vs Tofacitinib 5mg + csDMARD (Global Cohort); Test type: Non-Inferiority — Non-inferiority over tofacitinib on ACR20 was concluded if the lower limit of the multiplicity corrected 95% Confidence Interval (CI) in the difference in proportions (GSK3196165 minus tofacitinib) was greater than -12%; Regression, Logistic; Difference in proportion and 95% CI are generated from logistic regression model adjusted for Baseline TJC68, Baseline SJC66 and Treatment Group; Difference in Percentage = -14.7, 95% CI 2-sided [-21.3 to -8.1]
Statistical Analysis 2: Comparison: GSK3196165 150mg + csDMARD (Global Cohort) vs Tofacitinib 5mg + csDMARD (Global Cohort); Test type: Non-Inferiority — [test comment as in outcome 5, analysis 1]; Regression, Logistic; [statistical method as in outcome 5, analysis 1]; Difference in Percentage = -17.2, 95% CI 2-sided [-23.9 to -10.6]

6. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=10 (CDAI LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 32.8 | 34.3 | 49.6
  Week 52 | 38.3 | 38.0 | 56.8

7. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=10 (CDAI LDA) at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 6
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants in ITT set. Analysis was performed using multiple imputation method to handle missing data.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 37.5 | 15.9 | 46.4
  Week 52 | 40.2 | 38.2 | 41.3

8. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 12 (Global Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. CDAI remission is achieved when CDAI total score <=2.8. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 4.7 | 4.5 | 9.7 | 3.8

9. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. CDAI remission is achieved when CDAI total score <=2.8.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 6.9 | 7.2 | 17.9
  Week 52 | 11.9 | 10.8 | 21.2

10. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 9
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 6.6 | 5.7 | 11.0
  Week 52 | 11.4 | 5.6 | 17.2

11. Secondary Outcome: Percentage of Participants Achieving 50%/70% Improvement in American College of Rheumatology Criteria(ACR50/70) at Week 12 (Global Cohort)
Description: ACR50/70 is calculated as a 50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)]. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants
  ACR50 | 21.6 | 25.1 | 39.4 | 9.5
  ACR70 | 6.9 | 9.6 | 18.9 | 4.2

12. Secondary Outcome: Percentage of Participants Achieving ACR50/70 at Week 24 and ACR20/50/70 Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: ACR20/50/70 is calculated as a 20%/50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20%/50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)].
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  ACR20, Week 52 | 64.3 | 65.3 | 75.6
  ACR50, Week 24 | 31.6 | 32.8 | 53.6
  ACR50, Week 52 | 36.5 | 36.9 | 52.9
  ACR70, Week 24 | 14.0 | 13.0 | 28.7
  ACR70, Week 52 | 19.1 | 17.5 | 35.7

13. Secondary Outcome: Percentage of Participants Achieving ACR50/70 at Week 24 and ACR20/50/70 Week 52 for Placebo Switched Arms (Global Cohort)
Description: ACR20/50/70 is calculated as a 20%/50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)].
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  ACR20, Week 52 | 56.3 | 63.4 | 70.1
  ACR50, Week 24 | 35.6 | 27.6 | 41.8
  ACR50, Week 52 | 43.7 | 38.5 | 47.2
  ACR70, Week 24 | 18.7 | 10.5 | 21.8
  ACR70, Week 52 | 22.6 | 15.4 | 20.7

14. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score Using 28 Joint Count and C-Reactive Protein (DAS28-CRP) <=3.2 (DAS28-CRP LDA) at Week 12 (Global Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP greater than or equal to (<=)3.2. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 23.2 | 23.6 | 40.7 | 10.4

15. Secondary Outcome: Percentage of Participants Achieving DAS28 Erythrocyte Sedimentation Rate (ESR) <=3.2 (DAS28-ESR LDA) at Week 12 (Global Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in millimeter [mm]/hour[hr]), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 13.2 | 14.6 | 23.6 | 7.3

16. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP greater than or equal to (<=)3.2. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 31.3 | 33.0 | 55.3
  Week 52 | 35.4 | 36.4 | 53.9

17. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in millimeter [mm]/hour[hr]), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 19.9 | 24.1 | 37.1
  Week 52 | 26.2 | 22.9 | 38.8

18. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 16
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 37.5 | 19.3 | 42.7
  Week 52 | 41.4 | 31.4 | 39.6

19. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 17
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 30.2 | 14.2 | 23.4
  Week 52 | 28.0 | 16.6 | 31.5

20. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 12 (Global Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-CRP less than (<)2.6. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 11.5 | 12.0 | 23.2 | 5.5

21. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 12 (Global Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 7.1 | 6.1 | 12.6 | 3.8

22. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-CRP less than (<)2.6. A negative change from baseline in DAS28-CRP indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 16.7 | 19.6 | 38.0
  Week 52 | 23.6 | 21.2 | 41.2

23. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 8.7 | 11.7 | 23.4
  Week 52 | 14.3 | 11.7 | 19.9

24. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 22
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 23.3 | 11.5 | 23.8
  Week 52 | 30.4 | 19.8 | 26.4

25. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 23
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 13.4 | 6.2 | 13.4
  Week 52 | 16.1 | 11.5 | 13.4

26. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate (European League Against Rheumatism) EULAR Response at Week 12 (Global Cohort)
Description: DAS28-CRP and DAS28-ESR scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as; DAS28<=3.2 and DAS28 decrease from Baseline (>1.2: good response),(>0.6 to <=1.2: moderate response) and (<=0.6: no response); DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline (>1.2: moderate response),(>0.6 to <=1.2: moderate response) and (<=0.6: no response) and DAS28>5.1 and DAS28 decrease from Baseline (>1.2: moderate response),(>0.6 to <=1.2: no response) and (<=0.6: no response).If the post-Baseline DAS28-CRP score was missing, then the corresponding EULAR category was set to missing. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 70.0 | 71.3 | 83.8 | 46.3

27. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate EULAR Response at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: DAS28-CRP and DAS28-ESR scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as; if current DAS28 <=3.2 and DAS28 decrease from Baseline (>1.2: good response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response); if current DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response) and if current DAS28 >5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: no response) and (<=0.6: no response). If the post-Baseline DAS28-CRP score was missing, then the corresponding EULAR category was set to missing.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 79.8 | 80.5 | 90.4
  Week 52 | 80.3 | 78.9 | 88.4

28. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate EULAR Response at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 27
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 78.4 | 73.0 | 82.7
  Week 52 | 74.5 | 81.1 | 81.5

29. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 12 (Global Cohort)
Description: Boolean-based ACR/EULAR remission is achieved if all of the following requirements are met at the same timepoint: Tender Joint Count 68 (TJC68) <= 1, Swollen Joint Count 66 (SJC66) <= 1, high sensitivity C-reactive Protein (hsCRP) <= 1mg/dl and patient's global assessment of disease activity (PtGA) <= 10. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Week 12
Population: The analysis was performed on the ITT set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Participants | 13 | 12 | 15 | 3

30. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Boolean-based ACR/EULAR remission is achieved if all of the following requirements are met at the same timepoint: Tender Joint Count 68 (TJC68) <= 1, Swollen Joint Count 66 (SJC66) <= 1, high sensitivity C-reactive Protein (hsCRP) <= 1mg/dl and patient's global assessment of disease activity (PtGA) <= 10.
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 497 | 477 | 247
Participants
  Week 24 | 21 | 18 | 28
  Week 52: number analyzed (Participants) | 461 | 448 | 227
  Week 52 | 37 | 26 | 27

31. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 30
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants in ITT set. Only those participants with data available at the specified time points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 83 | 75 | 76
Participants
  Week 24 | 4 | 2 | 3
  Week 52: number analyzed (Participants) | 74 | 68 | 67
  Week 52 | 8 | 4 | 7

32. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression Van Der Heijde Modified Total Sharp Scores (mTSS) <= 0.5) at Week 12 (Global Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. No radiographic progression is defined as a change from Baseline in van der Heijde mTSS score of <=0.5. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms
Time Frame: Week 12
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Percentage of participants | 88.2 | 92.7 | 94.1 | 85.8

33. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression (mTSS <= 0.5) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. No radiographic progression is defined as a change from Baseline in van der Heijde mTSS score of <=0.5.
Time Frame: Week 24 and Week 52
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Percentage of participants
  Week 24 | 84.6 | 89.9 | 92.7
  Week 52 | 78.2 | 83.8 | 87.7

34. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression (mTSS <= 0.5) at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: as for outcome 33
Time Frame: Week 24 and Week 52
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Percentage of participants
  Week 24 | 88.1 | 82.2 | 83.9
  Week 52 | 85.6 | 71.9 | 87.9

35. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 12 (Global Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (PtGA and PhGA VAS with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Scores on a scale | -15.50 (0.680) | -16.31 (0.678) | -21.06 (0.878) | -9.56 (0.896)

36. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Baseline was defined as the latest pre-dose assessment with a non-missing value (NMV), including those from unscheduled visits. Change from Baseline (CB) was calculated by subtracting the post dose (PD) visit value from the Baseline value (BV).
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Scores on a scale
  Week 24 | -20.14 (0.669) | -20.68 (0.677) | -24.93 (0.848)
  Week 52 | -20.84 (0.750) | -21.14 (0.762) | -24.87 (0.936)

37. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Baseline was defined as the latest pre-dose assessment with a non-missing value (NMV), including those from unscheduled visits. Change from Baseline (CB) was calculated by subtracting the post dose (PD) visit value from the Baseline value (BV). For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Scores on a scale
  Week 24 | -20.26 (1.334) | -16.78 (1.396) | -20.60 (1.385)
  Week 52 | -20.52 (1.472) | -20.95 (1.547) | -22.01 (1.545)

38. Secondary Outcome: Change From Baseline in DAS28-CRP/DAS28-ESR at Week 12 (Global Cohort)
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in milimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value (NMV), including those from unscheduled visits. Change from Baseline (CB) was calculated by subtracting the post dose (PD) visit value from the Baseline value (BV).
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Scores on a scale
  DAS28-CRP | -1.28 (0.064) | -1.35 (0.064) | -2.02 (0.082) | -0.71 (0.085)
  DAS28-ESR | -1.34 (0.066) | -1.40 (0.066) | -1.95 (0.084) | -0.73 (0.087)

39. Secondary Outcome: Change From Baseline in DAS28-CRP/DAS28-ESR at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: as for outcome 38
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Scores on a scale
  DAS28-CRP, Week 24 | -1.65 (0.070) | -1.71 (0.071) | -2.45 (0.089)
  DAS28-CRP, Week 52 | -1.77 (0.079) | -1.76 (0.080) | -2.40 (0.098)
  DAS28-ESR, Week 24 | -1.73 (0.073) | -1.79 (0.074) | -2.40 (0.092)
  DAS28-ESR, Week 52 | -1.87 (0.084) | -1.82 (0.084) | -2.38 (0.102)

40. Secondary Outcome: Change From Baseline in DAS28-CRP/DAS28-ESR at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in milimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value (NMV), including those from unscheduled visits. Change from Baseline (CB) was calculated by subtracting the post dose (PD) visit value from the Baseline value (BV). For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Scores on a scale
  DAS28-CRP, Week 24 | -1.76 (0.139) | -1.39 (0.146) | -1.88 (0.145)
  DAS28-CRP, Week 52 | -1.81 (0.156) | -1.70 (0.164) | -1.97 (0.165)
  DAS28-ESR, Week 24 | -1.88 (0.144) | -1.48 (0.149) | -1.93 (0.148)
  DAS28-ESR, Week 52 | -1.88 (0.165) | -1.74 (0.172) | -1.96 (0.169)

41. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 12 (Global Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Scores on a scale | 0.31 (0.072) | 0.15 (0.073) | 0.09 (0.092) | 0.13 (0.095)

42. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score ranges from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Scores on a scale
  Week 24 | 0.42 (0.092) | 0.32 (0.094) | 0.15 (0.115)
  Week 52 | 0.84 (0.148) | 0.46 (0.150) | 0.30 (0.184)

43. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score ranges from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as the latest pre-dose assessment with a non-missing value (NMV), including those from unscheduled visits. Change from Baseline (CB) was calculated by subtracting the post dose (PD) visit value from the Baseline value (BV). For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Scores on a scale
  Week 24 | 0.18 (0.185) | 0.51 (0.196) | 0.21 (0.196)
  Week 52 | -0.05 (0.288) | 0.76 (0.304) | 0.09 (0.307)

44. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: HAQ-DI is a 20-question instrument that assesses the degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Scores on a scale
  Week 24 | -0.38 (0.033) | -0.37 (0.033) | -0.53 (0.041)
  Week 52 | -0.40 (0.035) | -0.37 (0.035) | -0.52 (0.043)

45. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: HAQ-DI is a 20-question instrument that assesses the degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value (NMV), including those from unscheduled visits. Change from Baseline (CB) was calculated by subtracting the post dose (PD) visit value from the Baseline value (BV). For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Scores on a scale
  Week 24 | -0.36 (0.065) | -0.38 (0.067) | -0.33 (0.067)
  Week 52 | -0.30 (0.069) | -0.37 (0.070) | -0.40 (0.071)

46. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 12 (Global Cohort)
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Scores on a scale | -18.06 (1.266) | -17.13 (1.256) | -27.17 (1.610) | -10.28 (1.657)

47. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Scores on a scale
  Week 24 | -23.32 (1.351) | -22.32 (1.371) | -31.27 (1.699)
  Week 52 | -25.42 (1.506) | -25.14 (1.525) | -31.49 (1.846)

48. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value (NMV), including those from unscheduled visits. Change from Baseline (CB) was calculated by subtracting the post dose (PD) visit value from the Baseline value (BV). For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1) and Week 24 and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Scores on a scale
  Week 24 | -23.26 (2.710) | -18.45 (2.793) | -22.88 (2.791)
  Week 52 | -23.71 (2.967) | -21.72 (3.071) | -21.62 (3.082)

49. Secondary Outcome: Change From Baseline in Short Form (SF)-36 Physical Component Scores at Week 12 (Global Cohort)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning(PF),bodily pain(BP),role limitations due to physical/emotional problems,general health(GH),mental health,social functioning,vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.PCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health.PCS is primarily derived from 4 domains(PF,role-physical,BP,GH) representing overall physical health.Positive change from baseline, reported using T-score change, indicates improvement in overall physical health.Quality Metric software was used for scoring.Baseline=latest pre-dose assessment with NMV, including those from unscheduled visits.CB=subtracting PD visit value from BV.For purpose of all analyses up to week12, placebo arms were pooled into single arm to primarily serve as reference for comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the ITT set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. For the purpose of all analyses up to week12, placebo arms were pooled into single placebo arm to primarily serve as reference for the comparison of active treatment arms. Analysis was performed using multiple imputation method to handle missing data.
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
T-Score | 4.29 (0.363) | 4.48 (0.361) | 6.58 (0.464) | 2.05 (0.478)

50. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores at Week 12 (Global Cohort)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning,bodily pain,role limitations due to physical/emotional problems,general health,mental health(MH),social functioning(SF),vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.MCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. MCS is primarily derived from 4 domains (SF,vitality,MH,role-emotional) representing overall mental health.Positive change from baseline, reported using T-score change, indicates improvement in overall mental health.Quality Metric software was used for scoring.Baseline=latest pre-dose assessment with NMV, including those from unscheduled visits.CB=subtracting PD visit value from BV.For purpose of all analyses up to week12, placebo arms were pooled into single arm to primarily serve as reference for comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 49
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
T-Score | 2.24 (0.474) | 2.68 (0.471) | 3.56 (0.604) | 2.21 (0.624)

51. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 12 (Global Cohort)
Description: Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning, bodily pain, role limitations due to physical and emotional problems, general health, mental health, social functioning, vitality. The MCS consists of 4 domains (social functioning, vitality, mental health, and role-emotional domains) and PCS consists of 4 domains (physical functioning, role-physical, bodily pain and general health). The individual question items are first summed for each item under the various sections. Then, those domain scores are weighted to a scale between 0 to 100, where higher score represents better health. A positive change from baseline indicates an improvement. Quality Metric software was used for scoring for SF-36. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the ITT set that includes all randomized participants who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. For the purpose of all analyses up to week12, placebo arms were pooled into single placebo arm to primarily serve as reference for the comparison of active treatment arms. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 506 | 514 | 252 | 244
Scores on a scale
  Bodily Pain | 14.82 (20.264) | 16.13 (20.997) | 23.75 (22.916) | 9.21 (21.040)
  General Health | 7.48 (16.025) | 6.74 (15.582) | 10.48 (15.647) | 5.16 (14.863)
  Mental Health | 6.21 (17.655) | 6.96 (18.312) | 9.13 (19.229) | 4.88 (18.257)
  Physical Function | 12.78 (19.321) | 14.47 (21.133) | 18.63 (20.724) | 8.42 (20.505)
  Role Emotional | 6.41 (24.390) | 7.90 (25.675) | 9.85 (24.815) | 7.00 (23.912)
  Role Physical | 12.08 (21.650) | 12.57 (22.044) | 17.66 (21.724) | 9.78 (20.593)
  Social Function | 8.10 (23.132) | 9.75 (25.484) | 14.78 (25.900) | 6.76 (23.984)
  Vitality | 8.99 (18.971) | 10.54 (19.349) | 15.18 (21.491) | 7.07 (18.624)

52. Secondary Outcome: Change From Baseline in SF-36 Physical Component Scores at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning(PF),bodily pain(BP),role limitations due to physical/emotional problems,general health(GH),mental health,social functioning,vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.PCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health.PCS is primarily derived from 4 domains(PF,role-physical,BP,GH) representing overall physical health.Positive change from baseline, reported using T-score change, indicates improvement in overall physical health.Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
T-Score
  Week 24 | 5.42 (0.416) | 5.24 (0.421) | 7.33 (0.520)
  Week 52 | 5.08 (0.460) | 5.06 (0.464) | 7.47 (0.569)

53. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning,bodily pain,role limitations due to physical/emotional problems,general health,mental health(MH),social functioning(SF),vitality.Each of 8 domains is scored using average, 0-100; higher score represents better health.MCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. MCS is primarily derived from 4 domains (SF,vitality,MH,role-emotional) representing overall mental health.Positive change from baseline, reported using T-score change, indicates improvement in overall mental health.Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
T-Score
  Week 24 | 2.69 (0.522) | 3.16 (0.528) | 4.80 (0.652)
  Week 52 | 3.06 (0.527) | 3.38 (0.530) | 4.08 (0.650)

54. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: as for outcome 51
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 494 | 486 | 249
Scores on a scale
  Bodily Pain, Week 24 | 18.06 (21.568) | 18.87 (23.164) | 26.26 (24.870)
  Bodily Pain, Week 52: number analyzed (Participants) | 461 | 459 | 234
  Bodily Pain, Week 52 | 19.38 (22.807) | 20.50 (23.781) | 27.01 (24.068)
  General Health, Week 24 | 8.80 (17.357) | 8.18 (16.569) | 11.82 (18.258)
  General Health, Week 52: number analyzed (Participants) | 461 | 459 | 234
  General Health, Week 52 | 8.72 (17.635) | 8.74 (17.157) | 12.71 (18.374)
  Mental Health, Week 24 | 7.33 (18.871) | 7.81 (19.930) | 11.24 (19.875)
  Mental Health, Week 52: number analyzed (Participants) | 461 | 459 | 234
  Mental Health, Week 52 | 8.03 (18.819) | 8.21 (19.132) | 9.87 (19.417)
  Physical Function, Week 24 | 16.20 (21.646) | 16.59 (22.660) | 21.73 (23.769)
  Physical Function, Week 52: number analyzed (Participants) | 461 | 459 | 234
  Physical Function, Week 52 | 16.90 (21.458) | 17.40 (23.162) | 22.31 (26.462)
  Role Emotional, Week 24 | 8.33 (27.318) | 10.01 (24.860) | 13.45 (24.656)
  Role Emotional, Week 52: number analyzed (Participants) | 461 | 459 | 234
  Role Emotional, Week 52 | 9.31 (24.987) | 10.77 (25.914) | 13.85 (25.643)
  Role Physical, Week 24 | 15.51 (22.052) | 15.60 (22.507) | 18.90 (22.618)
  Role Physical, Week 52: number analyzed (Participants) | 461 | 459 | 234
  Role Physical, Week 52 | 15.58 (23.558) | 16.29 (24.110) | 21.98 (24.671)
  Social Function, Week 24 | 10.25 (24.377) | 11.34 (26.893) | 15.91 (27.581)
  Social Function, Week 52: number analyzed (Participants) | 461 | 459 | 234
  Social Function, Week 52 | 11.23 (24.368) | 12.06 (26.941) | 14.42 (27.313)
  Vitality, Week 24 | 11.21 (20.320) | 12.71 (20.389) | 18.02 (22.463)
  Vitality, Week 52: number analyzed (Participants) | 461 | 459 | 234
  Vitality, Week 52 | 12.96 (20.197) | 12.58 (19.150) | 16.35 (22.327)

55. Secondary Outcome: Change From Baseline in SF-36 Physical Component Scores at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning(PF),bodily pain(BP),role limitations due to physical/emotional problems,general health(GH),mental health,social functioning,vitality. Each of 8 domains is scored using average, 0-100; higher score represents better health. PCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. PCS is primarily derived from 4 domains (PF,role-physical,BP,GH) representing overall physical health. Positive change from baseline, reported using T-score change, indicates improvement in overall physical health. Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
T-Score
  Week 24 | 5.89 (0.821) | 4.36 (0.851) | 5.43 (0.857)
  Week 52 | 4.15 (0.902) | 4.89 (0.929) | 3.99 (0.941)

56. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: SF-36 is health-related survey that assesses quality of life covering 8 domains:physical functioning,bodily pain,role limitations due to physical/emotional problems,general health,mental health(MH),social functioning(SF),vitality. Each of 8 domains is scored using average, 0-100; higher score represents better health. MCS was aggregated across the domains and scaled to T-score with mean of 50 and SD of 10; higher score represents better health. MCS is primarily derived from 4 domains (SF,vitality,MH,role-emotional) representing overall mental health. Positive change from baseline, reported using T-score change, indicates improvement in overall mental health. Quality Metric software was used for scoring. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: T-Score
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
T-Score
  Week 24 | 3.59 (1.041) | 4.37 (1.076) | 3.76 (1.082)
  Week 52 | 2.87 (1.051) | 4.53 (1.081) | 2.74 (1.092)

57. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: Short-Form 36 (SF-36) is a health-related survey that assesses quality of life covering 8 domains: physical functioning(PF), bodily pain(BP), role limitations due to physical and emotional problems, general health(GH), mental health(MH), social functioning(SF), vitality. The MCS consists of 4 domains (SF, vitality, MH, role-emotional) and PCS consists of 4 domains (PF, role-physical, BP, GH). The individual question items are first summed for each item under the various sections. Then, those domain scores are weighted to a scale between 0 to 100, where higher score represents better health. A positive change from baseline indicates an improvement. Quality Metric software was used for scoring for SF-36. Baseline was defined as latest pre-dose assessment with non-missing value, including from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: The analysis was performed on all randomized participants who switched from placebo to study intervention at Week 12. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 82 | 76 | 75
Scores on a scale
  Bodily Pain, Week 24 | 19.61 (22.430) | 17.93 (17.710) | 22.73 (21.012)
  Bodily Pain, Week 52: number analyzed (Participants) | 76 | 71 | 68
  Bodily Pain, Week 52 | 18.43 (23.444) | 19.35 (19.873) | 20.69 (23.501)
  General Health, Week 24 | 9.34 (13.259) | 8.96 (16.231) | 8.35 (17.087)
  General Health, Week 52: number analyzed (Participants) | 76 | 71 | 68
  General Health, Week 52 | 6.16 (15.885) | 10.52 (17.755) | 6.69 (16.707)
  Mental Health, Week 24 | 8.72 (19.623) | 10.20 (15.842) | 8.87 (19.270)
  Mental Health, Week 52: number analyzed (Participants) | 76 | 71 | 68
  Mental Health, Week 52 | 8.68 (19.585) | 12.25 (19.907) | 8.60 (19.256)
  Physical Function, Week 24 | 16.89 (20.407) | 17.30 (20.744) | 16.93 (21.433)
  Physical Function, Week 52: number analyzed (Participants) | 76 | 71 | 68
  Physical Function, Week 52 | 13.55 (24.025) | 19.72 (20.769) | 18.53 (20.608)
  Role Emotional, Week 24 | 9.35 (26.495) | 15.57 (25.325) | 11.44 (27.901)
  Role Emotional, Week 52: number analyzed (Participants) | 76 | 71 | 68
  Role Emotional, Week 52 | 6.91 (27.467) | 16.78 (28.189) | 10.29 (28.907)
  Role Physical, Week 24 | 16.92 (22.168) | 17.02 (19.568) | 20.17 (21.197)
  Role Physical, Week 52: number analyzed (Participants) | 76 | 71 | 68
  Role Physical, Week 52 | 14.80 (23.581) | 20.86 (20.727) | 17.46 (24.087)
  Social Function, Week 24 | 12.80 (25.381) | 12.17 (25.247) | 14.33 (24.634)
  Social Function, Week 52: number analyzed (Participants) | 76 | 71 | 68
  Social Function, Week 52 | 8.55 (29.312) | 16.20 (25.477) | 15.26 (24.131)
  Vitality, Week 24 | 14.25 (18.770) | 13.40 (18.839) | 13.67 (21.100)
  Vitality, Week 52: number analyzed (Participants) | 76 | 71 | 68
  Vitality, Week 52 | 13.32 (19.826) | 12.50 (21.417) | 11.31 (20.581)

58. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue at Week 12 (Global Cohort)
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271 | 270
Scores on a scale | 4.76 (0.482) | 4.91 (0.479) | 7.92 (0.615) | 3.68 (0.637)

59. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 271
Scores on a scale
  Week 24 | 6.10 (0.523) | 6.12 (0.528) | 8.37 (0.654)
  Week 52 | 6.97 (0.538) | 6.41 (0.543) | 8.38 (0.664)

60. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 91 | 89 | 90
Scores on a scale
  Week 24 | 6.95 (1.034) | 6.08 (1.072) | 6.87 (1.070)
  Week 52 | 5.73 (1.061) | 6.50 (1.096) | 6.01 (1.105)

61. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) (Global Cohort)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Fifteen participants in Placebo group received active treatment of Tofacitinib mistakenly from Week 4 instead of Week 12 as planned. They were added with the Tofacitinib arm in safety analysis.
Time Frame: Up to Week 59
Population: The analysis was performed on the Safety Set for Pooled Placebo (collected data till Week 12), GSK3196165 90 mg + MTX, GSK3196165 150 mg + MTX, Tofacitinib 5 mg + MTX (collected data till Week 59).
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 286 | 255
Participants
  Participants with AE | 420 | 408 | 224 | 127
  Participants with SAE | 44 | 43 | 31 | 6
  Participants with AESI | 72 | 75 | 32 | 5

62. Secondary Outcome: Change From Baseline in Hematology Parameter of White Blood Cell (WBC) Count, Platelet Count, Neutrophils, Lymphocytes at Week 12 (Giga Cells Per Liter) (Global Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters including WBC count, platelet count, neutrophils, lymphocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the Safety Set. Fifteen participants in Placebo group received active treatment of Tofacitinib mistakenly from Week 4 instead of Week 12 as planned. They were added with the Tofacitinib arm in safety analysis. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 494 | 490 | 267 | 229
Giga cells per liter (10^9/L)
  Lymphocytes: number analyzed (Participants) | 494 | 490 | 265 | 228
  Lymphocytes | 0.002 (0.5235) | -0.019 (0.5304) | 0.045 (0.5477) | -0.011 (0.4783)
  Neutrophils: number analyzed (Participants) | 494 | 490 | 265 | 228
  Neutrophils | -0.444 (1.8305) | -0.647 (1.9192) | -1.054 (2.1874) | 0.053 (1.9956)
  Platelets: number analyzed (Participants) | 484 | 486 | 264 | 225
  Platelets | -19.0 (50.74) | -19.9 (53.15) | -34.3 (64.33) | 0.8 (54.75)
  Leukocytes: number analyzed (Participants) | 492 | 488 | 267 | 229
  Leukocytes | -0.45 (1.919) | -0.70 (1.992) | -1.02 (2.215) | 0.02 (1.984)

63. Secondary Outcome: Change From Baseline in Hematology Parameter of WBC Count, Platelet Count, Neutrophils, Lymphocytes at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters including WBC count, platelet count, neutrophils, lymphocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: The analysis was performed on Safety Set. Fifteen participants in Placebo group received active treatment of Tofacitinib mistakenly from Week 4 instead of Week 12 as planned. They were added with the Tofacitinib arm in safety analysis. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 497 | 480 | 255
Giga cells per liter (10^9/L)
  Lymphocytes, Week 24 | 0.004 (0.5092) | -0.017 (0.5188) | 0.031 (0.5294)
  Lymphocytes, Week 52: number analyzed (Participants) | 416 | 410 | 215
  Lymphocytes, Week 52 | 0.001 (0.5679) | -0.012 (0.5487) | -0.143 (0.5739)
  Neutrophils, Week 24 | -0.508 (1.7714) | -0.647 (2.0762) | -1.135 (2.2376)
  Neutrophils, Week 52: number analyzed (Participants) | 416 | 410 | 215
  Neutrophils, Week 52 | -0.594 (1.8490) | -0.788 (2.1627) | -1.022 (2.4346)
  Platelets, Week 24: number analyzed (Participants) | 493 | 473 | 254
  Platelets, Week 24 | -16.4 (61.73) | -21.0 (56.36) | -32.0 (63.74)
  Platelets, Week 52: number analyzed (Participants) | 416 | 413 | 215
  Platelets, Week 52 | -24.9 (66.31) | -22.0 (63.94) | -37.6 (70.56)
  Leukocytes, Week 24: number analyzed (Participants) | 497 | 478 | 255
  Leukocytes, Week 24 | -0.50 (1.818) | -0.66 (2.129) | -1.17 (2.269)
  Leukocytes, Week 52: number analyzed (Participants) | 419 | 414 | 216
  Leukocytes, Week 52 | -0.59 (1.976) | -0.80 (2.346) | -1.22 (2.465)

64. Secondary Outcome: Change From Baseline in Hematology Parameter of WBC Count, Platelet Count, Neutrophils, Lymphocytes at Week 24 and Week 52 (Global Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters including WBC count, platelet count, neutrophils, lymphocytes. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: The analysis was performed on the Safety Set-Placebo switch. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 80 | 74 | 64
Giga cells per liter (10^9/L)
  Lymphocytes, Week 24 | -0.072 (0.4236) | 0.014 (0.5442) | -0.042 (0.5563)
  Lymphocytes, Week 52: number analyzed (Participants) | 72 | 67 | 56
  Lymphocytes, Week 52 | -0.085 (0.5077) | -0.071 (0.5098) | -0.243 (0.6030)
  Neutrophils, Week 24 | -0.582 (1.6685) | -0.255 (2.1106) | -0.745 (1.9306)
  Neutrophils, Week 52: number analyzed (Participants) | 72 | 67 | 56
  Neutrophils, Week 52 | -0.605 (1.8343) | -0.288 (2.2031) | -0.617 (2.1111)
  Platelets, Week 24: number analyzed (Participants) | 77 | 73 | 64
  Platelets, Week 24 | -11.6 (58.77) | -13.6 (40.78) | -36.1 (62.88)
  Platelets, Week 52: number analyzed (Participants) | 66 | 67 | 56
  Platelets, Week 52 | -17.8 (39.56) | -21.1 (44.72) | -27.8 (72.75)
  Leukocytes, Week 24: number analyzed (Participants) | 79 | 74 | 64
  Leukocytes, Week 24 | -0.64 (1.669) | -0.25 (2.204) | -0.84 (2.093)
  Leukocytes, Week 52: number analyzed (Participants) | 72 | 68 | 57
  Leukocytes, Week 52 | -0.65 (2.148) | -0.38 (2.259) | -0.94 (2.134)

65. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 12 (Global Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters hemoglobin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 492 | 489 | 267 | 231
Grams per liter (g/L) | 0.8 (7.50) | 0.1 (7.57) | 0.4 (8.53) | -1.0 (7.57)

66. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters hemoglobin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 497 | 479 | 255
Grams per liter (g/L)
  Week 24 | 0.5 (8.89) | 1.0 (8.57) | 1.9 (9.23)
  Week 52: number analyzed (Participants) | 421 | 416 | 218
  Week 52 | 0.6 (10.83) | 0.0 (10.12) | 1.0 (10.35)

67. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters hemoglobin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 79 | 74 | 64
Grams per liter (g/L)
  Week 24 | 1.2 (6.36) | 1.2 (6.10) | 3.2 (9.01)
  Week 52: number analyzed (Participants) | 72 | 68 | 57
  Week 52 | 0.8 (7.96) | 1.8 (8.99) | 2.1 (10.14)

68. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Gamma-Glutamyl Transpeptidase (GGT) at Week 12 (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameters including aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (AP) and gamma-glutamyl transferase (GGT) levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 511 | 504 | 273 | 231
International units per liter (IU/L)
  AP | -1.3 (19.79) | 0.4 (28.71) | -5.1 (19.95) | -1.6 (22.96)
  ALT: number analyzed (Participants) | 506 | 499 | 270 | 231
  ALT | 0.8 (14.14) | 1.2 (13.49) | 3.0 (15.73) | 0.3 (15.88)
  AST: number analyzed (Participants) | 509 | 504 | 272 | 230
  AST | 1.3 (8.34) | 2.0 (11.35) | 3.8 (12.23) | -0.1 (8.73)
  GGT | -1.5 (20.77) | 0.3 (44.60) | -1.1 (17.60) | -1.7 (25.38)

69. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of AST, ALT, AP, GGT at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameters including AST, ALT, AP and GGT levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 497 | 480 | 257
International units per liter (IU/L)
  AP, Week 24 | -0.3 (23.40) | 0.6 (20.47) | -7.9 (24.03)
  AP, Week 52: number analyzed (Participants) | 437 | 437 | 225
  AP, Week 52 | 0.3 (20.20) | 1.4 (22.40) | -5.1 (23.34)
  ALT, Week 24: number analyzed (Participants) | 496 | 477 | 256
  ALT, Week 24 | 1.0 (18.23) | 4.6 (63.38) | 4.1 (21.70)
  ALT, Week 52: number analyzed (Participants) | 432 | 426 | 222
  ALT, Week 52 | -0.1 (14.16) | 2.0 (16.35) | 3.7 (15.33)
  AST, Week 24: number analyzed (Participants) | 495 | 479 | 257
  AST, Week 24 | 1.2 (9.71) | 3.8 (45.20) | 4.2 (13.20)
  AST, Week 52: number analyzed (Participants) | 436 | 436 | 226
  AST, Week 52 | 1.0 (8.08) | 2.0 (11.47) | 3.9 (11.17)
  GGT, Week 24: number analyzed (Participants) | 497 | 479 | 257
  GGT, Week 24 | -1.2 (25.56) | 0.5 (32.53) | -1.6 (16.76)
  GGT, Week 52: number analyzed (Participants) | 437 | 437 | 226
  GGT, Week 52 | -1.0 (24.25) | 0.2 (22.40) | -0.1 (17.49)

70. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of AST, ALT, AP, GGT at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameters including AST, ALT, AP and GGT levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 83 | 74 | 64
International units per liter (IU/L)
  AP, Week 24 | -0.3 (15.77) | -3.5 (19.93) | -2.8 (23.41)
  AP, Week 52: number analyzed (Participants) | 72 | 69 | 58
  AP, Week 52 | -2.8 (19.07) | -1.6 (27.58) | -2.7 (26.76)
  ALT, Week 24: number analyzed (Participants) | 81 | 73 | 64
  ALT, Week 24 | -0.2 (14.86) | 0.2 (14.15) | 6.4 (15.92)
  ALT, Week 52: number analyzed (Participants) | 72 | 69 | 57
  ALT, Week 52 | 1.0 (20.01) | 0.7 (13.66) | 7.8 (24.01)
  AST, Week 24 | -0.2 (10.16) | 1.4 (6.42) | 5.0 (9.96)
  AST, Week 52: number analyzed (Participants) | 72 | 69 | 57
  AST, Week 52 | 1.3 (14.54) | 2.2 (7.07) | 7.0 (16.92)
  GGT, Week 24 | 0.8 (20.15) | -2.0 (18.05) | 0.0 (25.57)
  GGT, Week 52: number analyzed (Participants) | 72 | 69 | 58
  GGT, Week 52 | -2.1 (15.84) | -1.1 (16.29) | 0.8 (23.66)

71. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 12 (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameter total bilirubin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 506 | 499 | 271 | 231
Micromoles per liter (umol/L) | 0.3 (2.84) | 0.5 (2.68) | 0.5 (3.11) | 0.2 (2.78)

72. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameter total bilirubin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 496 | 477 | 256
Micromoles per liter (umol/L)
  Week 24 | 0.5 (2.66) | 0.5 (2.78) | 0.6 (2.73)
  Week 52: number analyzed (Participants) | 432 | 427 | 222
  Week 52 | 0.3 (2.66) | 0.6 (2.80) | 0.9 (2.83)

73. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameter total bilirubin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 81 | 73 | 64
Micromoles per liter (umol/L)
  Week 24 | 0.3 (3.07) | 0.3 (2.06) | 0.4 (2.79)
  Week 52: number analyzed (Participants) | 72 | 69 | 57
  Week 52 | -0.1 (2.88) | 0.6 (2.44) | 0.4 (2.20)

74. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 12 (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameter albumin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 511 | 504 | 273 | 231
Grams per liter (g/L) | 0.1 (2.56) | 0.1 (2.49) | 1.1 (2.60) | -0.3 (2.72)

75. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameter albumin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 497 | 479 | 257
Grams per liter (g/L)
  Week 24 | 0.2 (2.72) | 0.3 (2.59) | 1.6 (2.95)
  Week 52: number analyzed (Participants) | 437 | 437 | 227
  Week 52 | 0.3 (2.77) | 0.3 (2.88) | 1.3 (3.03)

76. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 24 and Week 52 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of clinical chemistry parameter albumin level. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 83 | 74 | 64
Grams per liter (g/L)
  Week 24 | 0.1 (2.33) | 0.6 (2.13) | 2.5 (2.99)
  Week 52: number analyzed (Participants) | 72 | 69 | 58
  Week 52 | -0.0 (2.87) | 0.9 (2.64) | 2.1 (3.22)

77. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 12 (Global Cohort)
Description: Blood samples were collected for the assessment of lipid profile of total cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: Blood samples were collected at indicated time points per schedule of assessment in protocol. Objectives and Endpoints section incorrectly states that Change from baseline in key laboratory parameters at Week 12 was a secondary objective, however for lipid panel, there is no corresponding time point in schedule of assessment. Consequently, the objective that can be assessed for the lipid panel is Week 4 and not Week 12 as no data collected. Week 4 is not pre-specified time point to report.
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0

78. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 24 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples were collected for the assessment of lipid profile of total cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: Blood samples were collected at indicated time points per schedule of assessment in protocol. Objectives and Endpoints section incorrectly states that Change from baseline in key laboratory parameters at Week 24 was a secondary objective, however for lipid panel, there is no corresponding time point in schedule of assessment. Consequently, the objective that can be assessed for the lipid panel is Week 16 and not Week 24 as no data collected. Week 16 is not pre-specified time point to report.
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0

79. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 24 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of lipid profile of total cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 78
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0

80. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: as for outcome 78
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 438 | 437 | 226
Millimoles per liter (mmol/L) | 0.121 (0.8198) | 0.129 (0.8076) | 0.402 (0.8794)

81. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 52 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of lipid profile of total cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For lipid profile assessments, baseline is interpreted as Week 4.
Time Frame: Baseline (Week 4) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 71 | 66 | 55
Millimoles per liter (mmol/L) | 0.198 (0.9586) | 0.255 (0.8086) | 0.691 (0.9233)

82. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Low-density Lipoprotein (LDL) Cholesterol, High-density Lipoprotein (HDL) Cholesterol at Week 12 (Global Cohort)
Description: Blood samples were collected for the assessment of fasting lipid profile including LDL cholesterol, HDL cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 77
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0

83. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 24 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples were collected for the assessment of fasting lipid profile including LDL cholesterol, HDL cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 78
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0

84. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 24 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of fasting lipid profile including LDL cholesterol, HDL cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 78
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0

85. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: as for outcome 83
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 438 | 437 | 226
Millimoles per liter (mmol/L)
  HDL Cholesterol, Direct | 0.026 (0.2415) | 0.010 (0.2812) | 0.157 (0.3184)
  LDL Cholesterol: number analyzed (Participants) | 432 | 436 | 226
  LDL Cholesterol | 0.076 (0.6971) | 0.093 (0.6396) | 0.191 (0.7423)

86. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 52 for Placebo Switched Arms (Global Cohort)
Description: Blood samples were collected for the assessment of fasting lipid profile including LDL cholesterol, HDL cholesterol levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For lipid profile assessments, baseline is interpreted as Week 4.
Time Frame: Baseline (Week 4) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 71 | 66 | 55
Millimoles per liter (mmol/L)
  HDL Cholesterol, Direct | -0.041 (0.2841) | 0.045 (0.2769) | 0.135 (0.3094)
  LDL Cholesterol: number analyzed (Participants) | 71 | 65 | 55
  LDL Cholesterol | 0.188 (0.7796) | 0.184 (0.6039) | 0.495 (0.7375)

87. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 12 (Global Cohort)
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 77
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0

88. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 24 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 78
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0

89. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 24 for Placebo Switched Arms (Global Cohort)
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 78
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 0 | 0 | 0

90. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Global Cohort)
Description: as for outcome 88
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 438 | 437 | 226
Millimoles per liter (mmol/L) | 0.045 (0.5902) | 0.054 (0.5970) | 0.117 (0.6444)

91. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 52 for Placebo Switched Arms (Global Cohort)
Description: TBlood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For lipid profile assessments, baseline is interpreted as Week 4.
Time Frame: Baseline (Week 4) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 71 | 66 | 55
Millimoles per liter (mmol/L) | 0.111 (0.4371) | 0.034 (0.5246) | 0.129 (0.5816)

92. Secondary Outcome: Number of Participants With National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE)>=Grade 3 Hematological/Clinical Chemistry Abnormalities (Global Cohort)
Description: Number of participants with NCI-CTCAE >=Grade 3 hematological/clinical chemistry abnormalities were summarized. Hematological and Clinical chemistry parameters were summarized according to the NCI-CTCAE, version 5.0: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling. Higher grade indicates more severity. Data is presented for only those parameters for which participants had worst case >=Grade 3 shifts from Baseline. Fifteen participants in Placebo group received active treatment of Tofacitinib mistakenly from Week 4 instead of Week 12 as planned. They were added with the Tofacitinib arm in safety analysis.
Time Frame: Up to Week 59
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 286 | 255
Participants
  Alanine aminotransferase increased,Total,Grade 3 | 4 | 5 | 4 | 1
  Aspartate aminotransferase increased,Total,Grade 3 | 2 | 3 | 1 | 1
  Anemia, Total, Grade 3 | 3 | 5 | 2 | 2
  Lymphocyte count decreased, Grade 3 | 9 | 11 | 9 | 3
  Neutrophil count decreased, Total, Grade 3 | 3 | 3 | 2 | 2
  Lymphocyte count decreased, Grade 4 | 0 | 0 | 9 | 0
  Hypertriglyceridemia, Total, Grade 3 | 10 | 0 | 2 | 0
  Aspartate aminotransferase increased, Total, Grade 4 | 0 | 2 | 0 | 0
  Alanine aminotransferase increased, Total, Grade 4 | 0 | 2 | 0 | 0
  Creatinine increased, Total, Grade 4 | 1 | 0 | 0 | 0
  Chronic Kidney Disease, Total, Grade 3 | 0 | 1 | 2 | 0
  Chronic Kidney Disease, Total, Grade 4 | 1 | 0 | 0 | 0
  Hemoglobin increased, Total, Grade 3 | 1 | 0 | 0 | 0
  White blood cell decreased, Total, Grade 3 | 2 | 0 | 0 | 0
  Neutrophil count decreased, Total, Grade 4 | 2 | 1 | 0 | 0
  Hypertriglyceridemia, Total, Grade 4 | 1 | 0 | 0 | 0

93. Secondary Outcome: Concentrations of Granulocyte-macrophage Colony Stimulating Factor (GM-CSF) Autoantibody (Global Cohort)
Description: Blood samples were collected for markers which may influence rheumatoid arthritis. Concentrations of GM-CSF autoantibodies was determined.
Time Frame: At baseline
Population: The analysis was performed on the Safety Set. Fifteen participants in Placebo group received active treatment of Tofacitinib mistakenly from Week 4 instead of Week 12 as planned. They were added with the Tofacitinib arm in safety analysis.
Measure: Mean (Standard Deviation); unit: Microgram per liter (ug/L)
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 286 | 91 | 89 | 75
Microgram per liter (ug/L) | 201.587 (519.9638) | 193.911 (402.0018) | 189.505 (344.7866) | 217.622 (399.6172) | 267.669 (642.5823) | 252.209 (671.7397)

94. Secondary Outcome: Number of Participants With Anti-GSK3196165 Antibodies (Global Cohort)
Description: Serum samples were collected for the determination of anti- GSK3196165 antibodies (ADA) using a validated electrochemiluminescence (ECL) immunoassay. The assay involved screening, confirmation and titration steps. If serum samples tested positive in the screening assay, they were considered 'potentially positive' and were further analyzed for the specificity using the confirmation assay. Samples that confirmed positive in the confirmation assay were reported as 'positive'. Confirmed positive ADA samples were further characterized in the titration assay to quasi-quantitate the amount of ADA in the sample. Additionally, confirmed positive ADA samples were also tested in a validated neutralizing antibody assay to determine the potential neutralizing activity of the ADA.
Time Frame: Up to Week 52
Population: as for outcome 93
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 545 | 539 | 286 | 91 | 89 | 75
Participants | 6 | 6 | 0 | 3 | 1 | 0

95. Secondary Outcome: Percentage of Participants Achieving Clinical Disease Activity Index (CDAI) Total Score Less Than or Equal to (<=)10 [CDAI Low Disease Activity (LDA)] at Week 12 (Asia Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Groups:
- GSK3196165 90mg + csDMARD (Asia Cohort): Participants in Asia Cohort received GSK3196165 90 mg subcutaneous (SC) injection once weekly for 52 weeks in combination with conventional synthetic disease-modifying antirheumatic drugs (csDMARD).
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 43 | 19 | 21
Percentage of participants | 13.0 | 12.0 | 58.0 | 19.0

96. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 (Asia Cohort)
Description: as for outcome 4
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 46 | 42 | 19 | 21
Scores on a scale | -0.22 (0.479) | -0.25 (0.537) | -0.47 (0.281) | 0.02 (0.577)

97. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=10 (CDAI LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Percentage of participants
  Week 24 | 21.0 | 19.0 | 53.0
  Week 52: number analyzed (Participants) | 31 | 32 | 15
  Week 52 | 45.0 | 41.0 | 47.0

98. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=10 (CDAI LDA) at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 97
Time Frame: Week 24 and Week 52
Population: The analysis was performed on all randomized participants who switched from placebo to study intervention at Week 12. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  Week 24 | 33.0 | 33.0 | 43.0
  Week 52: number analyzed (Participants) | 4 | 6 | 5
  Week 52 | 75.0 | 67.0 | 40.0

99. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 12 (Asia Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. CDAI remission is achieved when CDAI total score <=2.8. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: The analysis was performed on the ITT-Supplementary Asia Cohort Population, which consisted of participants randomized on or after 07-August-2021 who received at least one dose of study treatment. This population was based on the treatment the participant was randomized to. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 43 | 19 | 21
Percentage of participants | 2.0 | 0.0 | 11.0 | 0.0

100. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. CDAI remission is achieved when CDAI total score <=2.8. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Percentage of participants
  Week 24 | 0.0 | 7.0 | 24.0
  Week 52: number analyzed (Participants) | 31 | 32 | 15
  Week 52 | 6.0 | 16.0 | 13.0

101. Secondary Outcome: Percentage of Participants Achieving CDAI Total Score <=2.8 (CDAI Remission) at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 100
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  Week 24 | 0.0 | 0.0 | 0.0
  Week 52: number analyzed (Participants) | 4 | 6 | 5
  Week 52 | 25.0 | 0.0 | 20.0

102. Secondary Outcome: Percentage of Participants Achieving 50%/70% Improvement in American College of Rheumatology Criteria(ACR50/70) at Week 12 (Asia Cohort)
Description: ACR50/70 is calculated as a 50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)]. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 44 | 42 | 19 | 21
Percentage of participants
  ACR50 | 11.0 | 12.0 | 53.0 | 0.0
  ACR70 | 5.0 | 2.0 | 16.0 | 0.0

103. Secondary Outcome: Percentage of Participants Achieving ACR20/50/70 at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: ACR20/50/70 is calculated as a 20%/50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 20%/50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)]. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 37 | 42 | 17
Percentage of participants
  ACR20, Week 24 | 54.0 | 55.0 | 19.0
  ACR20, Week 52: number analyzed (Participants) | 30 | 31 | 15
  ACR20, Week 52 | 63.0 | 77.0 | 87.0
  ACR50, Week 24 | 19.0 | 24.0 | 53.0
  ACR50, Week 52: number analyzed (Participants) | 30 | 31 | 15
  ACR50, Week 52 | 37.0 | 48.0 | 53.0
  ACR70, Week 24 | 8.0 | 7.0 | 29.0
  ACR70, Week 52: number analyzed (Participants) | 30 | 31 | 15
  ACR70, Week 52 | 13.0 | 10.0 | 27.0

104. Secondary Outcome: Percentage of Participants Achieving ACR20/50/70 at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: ACR20/50/70 is calculated as a 20%/50%/70% improvement from Baseline in Tender Joint Count 68 (TJC68) and Swollen Joint Count 66 (SJC66) and a 50%/70% improvement in 3 of the following 5 measures: Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale (VAS) with values from 0=best to 100=worst), Physician Global Assessment of Arthritis Disease Activity (PhGA) [VAS with values from 0=best to 100=worst), Patient Assessment of Arthritis Pain (VAS with values from 0=no pain and 100=most severe pain), Health Assessment Questionnaire-Disability Index (HAQ-DI) (ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty) and an acute-phase reactant (high sensitivity C-reactive Protein mg/L (hsCRP)]. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  ACR20, Week 24 | 33.0 | 17.0 | 38.0
  ACR20, Week 52: number analyzed (Participants) | 4 | 6 | 6
  ACR20, Week 52 | 75.0 | 33.0 | 67.0
  ACR50, Week 24 | 0.0 | 0.0 | 43.0
  ACR50, Week 52: number analyzed (Participants) | 4 | 6 | 6
  ACR50, Week 52 | 50.0 | 17.0 | 67.0
  ACR70, Week 24 | 0.0 | 0.0 | 14.0
  ACR70, Week 52: number analyzed (Participants) | 4 | 6 | 6
  ACR70, Week 52 | 50.0 | 17.0 | 17.0

105. Secondary Outcome: Percentage of Participants Achieving Disease Activity Score Using 28 Joint Count and C-Reactive Protein (DAS28-CRP) <=3.2 (DAS28-CRP LDA) at Week 12 (Asia Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP greater than or equal to (<=)3.2. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 42 | 19 | 21
Percentage of participants | 16.0 | 21.0 | 58.0 | 10.0

106. Secondary Outcome: Percentage of Participants Achieving DAS28 Erythrocyte Sedimentation Rate (ESR) <=3.2 (DAS28-ESR LDA) at Week 12 (Asia Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in millimeter [mm]/hour[hr]), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 43 | 19 | 21
Percentage of participants | 20.0 | 9.0 | 47.0 | 10.0

107. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Low disease activity (LDA) is achieved when DAS28-CRP greater than or equal to (<=)3.2. A negative change from baseline in DAS28-CRP indicates an improvement. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Percentage of participants
  Week 24 | 24.0 | 21.0 | 53.0
  Week 52: number analyzed (Participants) | 31 | 32 | 15
  Week 52 | 39.0 | 34.0 | 67.0

108. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in millimeter [mm]/hour[hr]), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicate less disease activity. Low disease activity (LDA) is achieved when DAS28-ESR<=3.2. A negative change from baseline in DAS28-ESR indicates an improvement. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Percentage of participants
  Week 24 | 16.0 | 16.0 | 47.0
  Week 52: number analyzed (Participants) | 28 | 30 | 15
  Week 52 | 25.0 | 20.0 | 47.0

109. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <=3.2 (DAS28-CRP LDA) at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 107
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  Week 24 | 33.0 | 33.0 | 43.0
  Week 52: number analyzed (Participants) | 4 | 6 | 6
  Week 52 | 75.0 | 50.0 | 67.0

110. Secondary Outcome: Percentage of Participants Achieving DAS28-ESR <=3.2 (DAS28-ESR LDA) at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 108
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  Week 24 | 33.0 | 0.0 | 29.0
  Week 52: number analyzed (Participants) | 4 | 6 | 6
  Week 52 | 50.0 | 0.0 | 17.0

111. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 12 (Asia Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-CRP less than (<)2.6. A negative change from baseline in DAS28-CRP indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 42 | 19 | 21
Percentage of participants | 11.0 | 5.0 | 42.0 | 10.0

112. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 12 (Asia Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 43 | 19 | 21
Percentage of participants | 2.0 | 2.0 | 21.0 | 0.0

113. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: The DAS28-CRP is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), C-reactive protein (CRP) (in mg/L), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28- CRP scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-CRP less than (<)2.6. A negative change from baseline in DAS28-CRP indicates an improvement. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Percentage of participants
  Week 24 | 13.0 | 19.0 | 41.0
  Week 52: number analyzed (Participants) | 31 | 32 | 15
  Week 52 | 19.0 | 25.0 | 53.0

114. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: The DAS28-ESR is a measure of RA disease activity calculated using Tender Joint Count 28 (TJC28), Swollen Joint Count 28 (SJC28), Erythrocyte sedimentation rate (ESR) (in mm/hr), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst). DAS28-ESR scores range from 1.0 to 9.4, where lower scores indicates less disease activity. Remission is achieved when DAS28-ESR <2.6. A negative change from baseline in DAS28-ESR indicates an improvement. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Percentage of participants
  Week 24 | 8.0 | 12.0 | 29.0
  Week 52: number analyzed (Participants) | 28 | 30 | 15
  Week 52 | 7.0 | 17.0 | 20.0

115. Secondary Outcome: Percentage of Participants Achieving DAS28-CRP <2.6 (DAS28-CRP Remission) at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 113
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  Week 24 | 33.0 | 0.0 | 29.0
  Week 52: number analyzed (Participants) | 4 | 6 | 6
  Week 52 | 50.0 | 17.0 | 17.0

116. Secondary Outcome: Percentage of Participants Achieving DAS28 ESR <2.6 (DAS28-ESR Remission) at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 114
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  Week 24 | 0.0 | 0.0 | 0.0
  Week 52: number analyzed (Participants) | 4 | 6 | 6
  Week 52 | 25.0 | 0.0 | 17.0

117. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate European League Against Rheumatism (EULAR) Response at Week 12(Asia Cohort)
Description: DAS28-CRP and DAS28-ESR scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as; DAS28<=3.2 and DAS28 decrease from Baseline (>1.2: good response),(>0.6 to <=1.2: moderate response) and (<=0.6: no response); DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline (>1.2: moderate response),(>0.6 to <=1.2: moderate response) and (<=0.6: no response) and DAS28>5.1 and DAS28 decrease from Baseline (>1.2: moderate response),(>0.6 to <=1.2: no response) and (<=0.6: no response).If the post-Baseline DAS28-CRP score was missing, then the corresponding EULAR category was set to missing. Percentage values are rounded off.
Time Frame: Week 12
Population: The analysis was performed on the ITT-Supplementary Asia Cohort Population, which consisted of participants randomized on or after 07-August-2021 who received at least one dose of study treatment. Only those participants with data available at the indicated timepoints were analyzed. For the purpose of all analyses up to week 12, placebo arms were pooled into single placebo arm to primarily serve as reference for comparison of active treatment arms.
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 44 | 41 | 19 | 21
Percentage of participants | 66.0 | 61.0 | 84.0 | 33.0

118. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate EULAR Response at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: DAS28-CRP and DAS28-ESR scores were categorized using EULAR response criteria. Response at a given time point was defined based on the combination of current DAS28 score and the improvement in the current DAS28 score relative to Baseline. The definition of no response, moderate response and good response was as; if current DAS28 <=3.2 and DAS28 decrease from Baseline (>1.2: good response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response); if current DAS28 >3.2 to <=5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: moderate response) and (<=0.6: no response) and if current DAS28 >5.1 and DAS28 decrease from Baseline value (>1.2: moderate response), (>0.6 to <=1.2: no response) and (<=0.6: no response). If the post-Baseline DAS28-CRP score was missing, then the corresponding EULAR category was set to missing. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 37 | 42 | 17
Percentage of participants
  Week 24 | 65.0 | 64.0 | 94.0
  Week 52: number analyzed (Participants) | 30 | 31 | 15
  Week 52 | 70.0 | 84.0 | 100.0

119. Secondary Outcome: Percentage of Participants Achieving a Good/Moderate EULAR Response at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 118
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Percentage of participants
  Week 24 | 50.0 | 50.0 | 100.0
  Week 52: number analyzed (Participants) | 4 | 6 | 6
  Week 52 | 100.0 | 100.0 | 100.0

120. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 12 (Asia Cohort)
Description: as for outcome 29
Time Frame: Week 12
Population: The analysis was performed on the ITT-Supplementary Asia Cohort Population, which consisted of participants randomized on or after 07-August-2021 who received at least one dose of study treatment. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 42 | 19 | 21
Participants | 1 | 0 | 1 | 0

121. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 30
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Participants
  Week 24 | 0 | 0 | 3
  Week 52: number analyzed (Participants) | 31 | 32 | 15
  Week 52 | 0 | 2 | 2

122. Secondary Outcome: Number of Participants Achieving ACR/EULAR Remission at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 30
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Participants
  Week 24 | 0 | 0 | 1
  Week 52: number analyzed (Participants) | 4 | 6 | 6
  Week 52 | 0 | 0 | 0

123. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression Van Der Heijde Modified Total Sharp Scores (mTSS) <= 0.5) at Week 12 (Asia Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. No radiographic progression is defined as a change from Baseline in van der Heijde mTSS score of <=0.5. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms. Percentage values are rounded off.
Time Frame: Week 12
Population: as for outcome 99
Measure: Number; unit: Percentage of participants
Groups:
- Pooled Placebo (Asia Cohort): Participants from Asia cohort received Placebo weekly SC injection in combination with csDMARD until Week 12. The placebo arms are pooled into a single placebo arm.
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 9 | 6 | 3 | 2
Percentage of participants | 67.0 | 67.0 | 67.0 | 100.0

124. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression (mTSS <= 0.5) at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. No radiographic progression is defined as a change from Baseline in van der Heijde mTSS score of <=0.5. Percentage values are rounded off.
Time Frame: Week 24 and Week 52
Population: as for outcome 97
Measure: Number; unit: Percentage of participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 5 | 2
Percentage of participants
  Week 24 | 83.0 | 60.0 | 50.0
  Week 52: number analyzed (Participants) | 5 | 3 | 2
  Week 52 | 40.0 | 100.0 | 50.0

125. Secondary Outcome: Percentage of Participants Achieving no Radiographic Progression (mTSS <= 0.5) at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 124
Time Frame: Week 24 and Week 52
Population: as for outcome 98
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 1 | 1 | 0
Percentage of participants
  Week 24 | 100.0 | 100.0 |
  Week 52 | 100.0 | 100.0 |

126. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 12 (Asia Cohort)
Description: as for outcome 35
Time Frame: Baseline (Day 1) and week 12
Population: as for outcome 99
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 44 | 42 | 19 | 21
Scores on a scale | -13.75 (10.935) | -10.91 (11.649) | -19.47 (12.718) | -4.38 (8.640)

127. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Clinical Disease Activity Index (CDAI) total score is a composite score consisting of the sum of Swollen Joint Count 28 (TJC28), Tender Joint Count 28 (TJC28), Patient's Global Assessment of Arthritis Disease Activity (PtGA) (visual analogue scale with values from 0=best to 100=worst) and Physician Global Assessment of Arthritis Disease Activity (PhGA) (visual analogue scale with values from 0=best to 100=worst). PtGA and PhGA are transformed to a 0-10 scale before computing the CDAI total score. CDAI total score ranges from 0 to 76 with higher values representing higher disease activity. Low disease activity (LDA) is achieved when CDAI total score <=10. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 37 | 42 | 17
Scores on a scale
  Week 24 | -15.27 (12.329) | -13.39 (10.575) | -21.44 (11.208)
  Week 52: number analyzed (Participants) | 30 | 31 | 15
  Week 52 | -18.29 (13.199) | -19.35 (13.923) | -23.21 (12.303)

128. Secondary Outcome: Change From Baseline in CDAI Total Score at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 37
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Scores on a scale
  Week 24 | -8.78 (6.086) | -12.28 (10.842) | -20.47 (12.133)
  Week 52: number analyzed (Participants) | 4 | 6 | 5
  Week 52 | -16.28 (5.351) | -17.47 (11.166) | -23.18 (13.070)

129. Secondary Outcome: Change From Baseline in DAS28-CRP and DAS28-ESR at Week 12 (Asia Cohort)
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in milimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 99
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 44 | 42 | 19 | 21
Scores on a scale
  DAS28-CRP: number analyzed (Participants) | 44 | 41 | 19 | 21
  DAS28-CRP | -1.26 (1.034) | -1.05 (0.968) | -2.27 (1.089) | -0.47 (0.950)
  DAS28-ESR | -1.33 (1.023) | -1.11 (0.964) | -2.15 (1.161) | -0.40 (0.937)

130. Secondary Outcome: Change From Baseline in DAS28-CRP and DAS28-ESR at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in milimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 37 | 42 | 17
Scores on a scale
  DAS28-CRP, Week 24 | -1.41 (1.221) | -1.28 (1.086) | -2.29 (1.037)
  DAS28-CRP, Week 52: number analyzed (Participants) | 30 | 31 | 15
  DAS28-CRP, Week 52 | -1.63 (1.353) | -1.82 (1.262) | -2.47 (1.253)
  DAS28-ESR, Week 24 | -1.50 (1.153) | -1.27 (1.121) | -2.30 (1.246)
  DAS28-ESR, Week 52: number analyzed (Participants) | 28 | 29 | 15
  DAS28-ESR, Week 52 | -1.76 (1.358) | -1.84 (1.303) | -2.42 (1.318)

131. Secondary Outcome: Change From Baseline in DAS28-CRP/DAS28-ESR at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: DAS28-CRP and DAS28-ESR are measure of RA disease activity calculated using Swollen Joint Count 28 (SJC28), Tender Joint Count 28 (TJC28), high sensitivity C-reactive Protein (hsCRP in mg/L)/Erythrocyte sedimentation rate (ESR) [ESR in milimeter/hour (mm/hr)] and patient's global assessment of disease activity (PtGA) transformed to a 0-10 scale. Total score approximate range 0-9.4, with higher scores indicating more disease activity. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Scores on a scale
  DAS28-CRP, Week 24 | -1.27 (1.171) | -1.08 (0.852) | -2.14 (1.242)
  DAS28-CRP, Week 52: number analyzed (Participants) | 4 | 6 | 6
  DAS28-CRP, Week 52 | -2.24 (1.200) | -1.52 (1.005) | -2.63 (1.244)
  DAS28-ESR, Week 24 | -0.91 (1.216) | -0.99 (0.897) | -2.06 (1.053)
  DAS28-ESR, Week 52: number analyzed (Participants) | 4 | 6 | 6
  DAS28-ESR, Week 52 | -1.82 (1.183) | -1.46 (0.912) | -2.48 (1.186)

132. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 12 (Asia Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 99
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 9 | 6 | 3 | 2
Scores on a scale | 1.22 (2.476) | 3.42 (7.889) | 0.33 (0.577) | 0.25 (0.354)

133. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 5 | 2
Scores on a scale
  Week 24 | -0.08 (0.665) | 5.60 (10.922) | 0.50 (0.707)
  Week 52: number analyzed (Participants) | 5 | 3 | 2
  Week 52 | 1.40 (1.673) | 0.00 (0.000) | 0.50 (0.707)

134. Secondary Outcome: Change From Baseline in Van Der Heijde mTSS at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: Van der Heijde mTSS is utilized for scoring radiographs of hands and feet in rheumatoid arthritis. This method includes 16 areas of erosions, and 15 areas for joint space narrowing (JSN) in each hand, and 6 areas for erosions and 6 areas JSN in each foot. The total mTSS score is the sum of erosion (maximum of 280) and JSN (maximum of 168) scores. The score range from 0 to 448 for mTSS with higher values representing higher disease activity. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1. NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 1 | 1 | 0
Scores on a scale
  Week 24 | 0.50 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived. | 0.00 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived. |
  Week 52 | 0.50 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived. | 0.00 (NA) — NA indicate data not available since only one participant was analyzed, therefore standard deviation was not derived. |

135. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: HAQ-DI is a 20-question instrument that assesses the degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 42 | 17
Scores on a scale
  HAQ-Disability Index, Week 24 | -0.25 (0.569) | -0.29 (0.524) | -0.48 (0.266)
  HAQ-Disability Index, Week 52: number analyzed (Participants) | 32 | 31 | 15
  HAQ-Disability Index, Week 52 | -0.36 (0.573) | -0.40 (0.604) | -0.59 (0.483)

136. Secondary Outcome: Change From Baseline in HAQ-DI at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: HAQ-DI is a 20-question instrument that assesses the degree of difficulty of a participant in accomplishing tasks in eight functional areas: dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Overall HAQ-DI score was computed as sum of the domain scores divided by the number of domains answered. The total possible score ranges from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. A negative change from baseline indicates an improvement. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Scores on a scale
  HAQ-Disability Index, Week 24 | -0.33 (0.921) | -0.02 (0.436) | -0.46 (0.431)
  HAQ-Disability Index, Week 52: number analyzed (Participants) | 4 | 6 | 7
  HAQ-Disability Index, Week 52 | -0.19 (1.139) | -0.19 (0.438) | -0.52 (0.442)

137. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 12 (Asia Cohort)
Description: as for outcome 46
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 99
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 46 | 42 | 19 | 21
Scores on a scale | -20.0 (22.57) | -18.0 (25.37) | -21.2 (22.91) | -1.8 (21.00)

138. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 47
Time Frame: Baseline (Day 1) and Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 42 | 17
Scores on a scale
  Week 24 | -24.4 (22.90) | -25.2 (25.71) | -32.9 (25.97)
  Week 52: number analyzed (Participants) | 32 | 31 | 15
  Week 52 | -30.4 (26.98) | -27.9 (23.51) | -33.0 (23.04)

139. Secondary Outcome: Change From Baseline in Arthritis Pain VAS at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: For the Arthritis Pain VAS, participants assess the severity of their current arthritis pain using a continuous visual analogue scale (VAS) with anchors at "0" (no pain) and "100" (most severe pain). A negative change from baseline indicates an improvement. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1) and Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Scores on a scale
  Week 24 | -14.2 (20.71) | -13.5 (27.57) | -27.0 (21.86)
  Week 52: number analyzed (Participants) | 4 | 6 | 7
  Week 52 | -32.3 (14.45) | -21.8 (34.17) | -34.4 (27.50)

140. Secondary Outcome: Change From Baseline in Short Form (SF)-36 Physical Component Scores at Week 12 (Asia Cohort)
Description: as for outcome 49
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the ITT-Supplementary Asia Cohort Population, which consisted of participants randomized on or after 07-August-2021 who received at least one dose of study treatment. Only those participants with data available at the indicated timepoints were analyzed. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 42 | 19 | 21
T-Score | 4.051 (6.1927) | 3.040 (5.8359) | 8.312 (6.6143) | 0.222 (4.5222)

141. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores at Week 12 (Asia Cohort)
Description: as for outcome 50
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 42 | 19 | 21
T-Score | 1.529 (9.2379) | 2.197 (8.4871) | 1.149 (7.6184) | 0.392 (7.0528)

142. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 12 (Asia Cohort)
Description: as for outcome 51
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 140
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 42 | 19 | 21
Scores on a scale
  Bodily Pain | 12.64 (13.888) | 7.93 (14.984) | 23.42 (22.741) | 1.62 (18.712)
  General Health | 6.33 (17.092) | 2.86 (13.448) | 9.16 (15.174) | -4.05 (14.928)
  Mental Health | 4.00 (17.340) | 1.43 (14.579) | 1.32 (14.419) | 0.24 (13.179)
  Physical Function | 8.67 (15.537) | 8.10 (17.355) | 14.74 (19.037) | 1.90 (18.740)
  Role Emotional | 5.93 (20.150) | 7.54 (23.268) | 7.89 (21.957) | 2.38 (25.020)
  Role Physical | 8.89 (16.722) | 8.33 (23.494) | 20.07 (30.730) | 2.98 (19.924)
  Social Function | 3.06 (20.670) | 8.63 (20.379) | 13.82 (19.937) | 0.00 (16.298)
  Vitality | 7.22 (20.684) | 8.48 (15.849) | 9.54 (20.023) | 2.08 (11.238)

143. Secondary Outcome: Change From Baseline in SF-36 Physical Component Scores at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 52
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 37 | 42 | 17
T-Score
  Week 24 | 4.220 (7.5564) | 3.362 (5.9357) | 7.826 (9.0545)
  Week 52: number analyzed (Participants) | 31 | 31 | 15
  Week 52 | 4.646 (6.7378) | 5.328 (5.8824) | 9.942 (5.7938)

144. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 53
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 37 | 42 | 17
T-Score
  Week 24 | -0.157 (8.7537) | 2.741 (6.6865) | 0.071 (8.0170)
  Week 52: number analyzed (Participants) | 31 | 31 | 15
  Week 52 | 3.837 (9.6474) | 0.918 (10.3466) | 1.923 (9.4063)

145. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 51
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 37 | 42 | 17
Scores on a scale
  Bodily Pain, Week 24 | 13.43 (18.292) | 8.88 (13.862) | 30.59 (25.048)
  Bodily Pain, Week 52: number analyzed (Participants) | 31 | 31 | 15
  Bodily Pain, Week 52 | 16.77 (17.333) | 16.97 (16.956) | 30.20 (23.035)
  General Health, Week 24 | 4.97 (19.591) | 4.19 (14.101) | 2.41 (12.037)
  General Health, Week 52: number analyzed (Participants) | 31 | 31 | 15
  General Health, Week 52 | 5.74 (17.216) | 4.13 (14.509) | 10.87 (13.958)
  Mental Health, Week 24 | 0.68 (18.226) | 4.17 (13.521) | 2.65 (9.701)
  Mental Health, Week 52: number analyzed (Participants) | 31 | 31 | 15
  Mental Health, Week 52 | 7.42 (18.343) | 1.29 (17.510) | 6.00 (17.341)
  Physical Function, Week 24 | 6.08 (18.264) | 10.60 (17.916) | 14.71 (20.269)
  Physical Function, Week 52: number analyzed (Participants) | 31 | 31 | 15
  Physical Function, Week 52 | 10.00 (17.512) | 11.29 (17.367) | 21.67 (17.491)
  Role Emotional, Week 24 | 1.58 (22.209) | 8.53 (19.259) | 9.80 (25.215)
  Role Emotional, Week 52: number analyzed (Participants) | 31 | 31 | 15
  Role Emotional, Week 52 | 9.41 (20.609) | 8.87 (23.267) | 11.11 (21.973)
  Role Physical, Week 24 | 8.45 (24.572) | 8.63 (20.332) | 18.01 (40.437)
  Role Physical, Week 52: number analyzed (Participants) | 31 | 31 | 15
  Role Physical, Week 52 | 13.31 (18.381) | 12.90 (23.768) | 21.67 (30.969)
  Social Function, Week 24 | 2.70 (18.194) | 8.63 (16.904) | 3.68 (37.699)
  Social Function, Week 52: number analyzed (Participants) | 31 | 31 | 15
  Social Function, Week 52 | 10.48 (20.941) | 5.24 (22.770) | 11.67 (28.530)
  Vitality, Week 24 | 5.07 (22.040) | 8.04 (15.937) | 4.78 (25.342)
  Vitality, Week 52: number analyzed (Participants) | 31 | 31 | 15
  Vitality, Week 52 | 11.49 (22.308) | 6.05 (21.377) | 11.25 (23.170)

146. Secondary Outcome: Change From Baseline in SF-36 Physical Component Scores at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 55
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
T-Score
  Week 24 | 1.762 (5.8183) | 1.675 (6.9009) | 5.544 (5.4800)
  Week 52: number analyzed (Participants) | 4 | 6 | 7
  Week 52 | 3.818 (3.4904) | 3.268 (4.8182) | 7.024 (6.0185)

147. Secondary Outcome: Change From Baseline in SF-36 Mental Component Scores at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 56
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
T-Score
  Week 24 | 3.158 (8.1659) | 3.950 (5.3971) | 4.889 (8.1905)
  Week 52: number analyzed (Participants) | 4 | 6 | 7
  Week 52 | -0.028 (9.4600) | -1.940 (8.3373) | 2.401 (6.1426)

148. Secondary Outcome: Change From Baseline in SF-36 Domain Scores at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 57
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Scores on a scale
  Bodily Pain, Week 24 | 18.83 (23.017) | 12.17 (26.180) | 18.00 (23.951)
  Bodily Pain, Week 52: number analyzed (Participants) | 4 | 6 | 7
  Bodily Pain, Week 52 | 13.50 (26.889) | 12.83 (37.280) | 23.00 (20.905)
  General Health, Week 24 | -3.83 (14.689) | 0.83 (16.558) | -1.29 (12.148)
  General Health, Week 52: number analyzed (Participants) | 4 | 6 | 7
  General Health, Week 52 | 5.00 (14.697) | -0.83 (13.934) | 0.57 (18.911)
  Mental Health, Week 24 | 9.17 (13.197) | 5.83 (12.813) | 14.29 (5.345)
  Mental Health, Week 52: number analyzed (Participants) | 4 | 6 | 7
  Mental Health, Week 52 | 1.25 (13.769) | -2.50 (16.355) | 6.43 (7.480)
  Physical Function, Week 24 | 0.01 (17.887) | 2.50 (15.732) | 25.71 (18.356)
  Physical Function, Week 52: number analyzed (Participants) | 4 | 6 | 7
  Physical Function, Week 52 | 2.51 (18.925) | 5.83 (10.205) | 21.43 (15.738)
  Role Emotional, Week 24 | 11.11 (24.532) | 9.72 (16.171) | 15.48 (40.379)
  Role Emotional, Week 52: number analyzed (Participants) | 4 | 6 | 7
  Role Emotional, Week 52 | 0.00 (11.785) | -2.78 (21.515) | 11.91 (27.154)
  Role Physical, Week 24 | 13.54 (15.520) | 7.29 (10.013) | 15.18 (21.907)
  Role Physical, Week 52: number analyzed (Participants) | 4 | 6 | 7
  Role Physical, Week 52 | 9.38 (14.878) | 1.04 (14.479) | 16.96 (25.697)
  Social Function, Week 24 | -2.08 (20.026) | 4.17 (6.455) | 3.57 (17.252)
  Social Function, Week 52: number analyzed (Participants) | 4 | 6 | 7
  Social Function, Week 52 | 3.13 (31.250) | -6.25 (15.309) | 10.71 (18.298)
  Vitality, Week 24 | 3.13 (11.693) | 11.46 (14.479) | 15.18 (8.733)
  Vitality, Week 52: number analyzed (Participants) | 4 | 6 | 7
  Vitality, Week 52 | 4.69 (23.593) | 8.33 (6.455) | 8.93 (14.815)

149. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue at Week 12 (Asia Cohort)
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 99
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 46 | 42 | 19 | 21
Scores on a scale | 2.4 (8.01) | 4.0 (6.58) | 6.4 (7.64) | 0.3 (9.00)

150. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 97
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 42 | 17
Scores on a scale
  Week 24 | 1.9 (9.22) | 4.7 (5.96) | 5.1 (10.18)
  Week 52: number analyzed (Participants) | 32 | 31 | 15
  Week 52 | 3.3 (8.91) | 5.3 (7.65) | 7.7 (8.91)

151. Secondary Outcome: Change From Baseline in FACIT-Fatigue at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: The Functional Assessment of Chronic Illness Therapy (FACIT)-fatigue is a validated patient-reported measure of 13 statements regarding the feeling of fatigue. The total score ranges from 0 to 52 with higher values representing a lower fatigue and a better quality of life. A positive change from baseline in FACIT-fatigue indicates an improvement. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For efficacy assessments baseline is interpreted as Day 1.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 98
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Scores on a scale
  Week 24 | 6.3 (5.16) | 1.3 (4.93) | 3.0 (10.17)
  Week 52: number analyzed (Participants) | 4 | 6 | 7
  Week 52 | 4.0 (6.16) | 2.2 (1.94) | 2.0 (7.94)

152. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) (Asia Cohort)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. A SAE is any untoward medical occurrence that, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity and/or can result in death.
Time Frame: Up to Week 59
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo (Asian Cohort): Participants received Placebo weekly SC injection in combination with csDMARD until Week 12. The placebo arms are pooled into a single placebo arm.
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asian Cohort)
Number analyzed (Participants) | 47 | 49 | 19 | 23
Participants
  AE | 37 | 43 | 18 | 14
  SAE | 5 | 4 | 2 | 1
  AESI | 4 | 6 | 2 | 0

153. Secondary Outcome: Change From Baseline in Hematology Parameter of White Blood Cell (WBC) Count, Platelet Count, Neutrophils, Lymphocytes at Week 12 (Giga Cells Per Liter) (Asia Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters including WBC count, platelet count, neutrophils, lymphocytes. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: The analysis was performed on the Safety Set. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 43 | 19 | 21
Giga cells per liter (10^9/L)
  WBC count | -0.48 (1.369) | -0.35 (1.699) | -1.25 (1.038) | -0.18 (1.518)
  Platelet count | -17.8 (51.99) | -20.4 (44.57) | -22.9 (50.17) | 5.7 (48.47)
  Neutrophils | -0.654 (1.3274) | -0.473 (1.5847) | -1.316 (1.0213) | -0.352 (1.2533)
  Lymphocytes | 0.094 (0.3241) | 0.069 (0.3391) | 0.070 (0.3942) | 0.117 (0.4069)

154. Secondary Outcome: Change From Baseline in Hematology Parameter of WBC Count, Platelet Count, Neutrophils, Lymphocytes at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters including WBC count, platelet count, neutrophils, lymphocytes. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: The analysis was performed on Safety Set participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Giga cells per liter (10^9/L)
  WBC count, Week 24 | -0.42 (1.780) | -0.56 (1.467) | -0.26 (3.492)
  WBC count, Week 52: number analyzed (Participants) | 29 | 28 | 16
  WBC count, Week 52 | -0.60 (1.538) | -0.50 (1.338) | -1.30 (1.207)
  Platelet count, Week 24 | -24.8 (61.57) | -8.0 (39.63) | -3.2 (74.58)
  Platelet count, Week 52: number analyzed (Participants) | 29 | 28 | 16
  Platelet count, Week 52 | -27.4 (54.86) | -24.5 (53.19) | -28.6 (51.39)
  Neutrophils, Week 24 | -0.632 (1.7911) | -0.737 (1.3842) | -0.829 (1.7091)
  Neutrophils, Week 52: number analyzed (Participants) | 29 | 28 | 16
  Neutrophils, Week 52 | -0.794 (1.6493) | -0.475 (1.1881) | -0.828 (1.2338)
  Lymphocytes, Week 24 | 0.107 (0.3436) | 0.114 (0.2605) | 0.454 (1.7675)
  Lymphocytes, Week 52: number analyzed (Participants) | 29 | 28 | 16
  Lymphocytes, Week 52 | 0.129 (0.3706) | -0.002 (0.2894) | -0.414 (0.3126)

155. Secondary Outcome: Change From Baseline in Hematology Parameter of WBC Count, Platelet Count, Neutrophils, Lymphocytes at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: Blood samples were collected for the assessment of change from baseline in hematology parameters including WBC count, platelet count, neutrophils, lymphocytes. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Giga cells per liter (10^9/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Giga cells per liter (10^9/L)
  WBC count, Week 24 | -0.10 (1.404) | -1.10 (0.729) | -0.53 (1.559)
  WBC count, Week 52: number analyzed (Participants) | 4 | 5 | 6
  WBC count, Week 52 | -0.28 (0.544) | -0.08 (1.057) | 0.85 (1.285)
  Platelet count, Week 24 | -33.5 (39.29) | 1.2 (45.66) | -54.4 (72.52)
  Platelet count, Week 52: number analyzed (Participants) | 4 | 5 | 6
  Platelet count, Week 52 | -33.8 (48.88) | -27.4 (49.23) | -62.7 (67.67)
  Neutrophils, Week 24 | 0.042 (1.1970) | -1.153 (0.8378) | -0.599 (1.6470)
  Neutrophils, Week 52: number analyzed (Participants) | 4 | 5 | 6
  Neutrophils, Week 52 | -0.205 (0.3770) | -0.040 (0.6118) | 1.305 (1.0918)
  Lymphocytes, Week 24 | -0.160 (0.2929) | 0.185 (0.3747) | 0.030 (0.4946)
  Lymphocytes, Week 52: number analyzed (Participants) | 4 | 5 | 6
  Lymphocytes, Week 52 | 0.093 (0.1962) | 0.092 (0.3667) | -0.568 (0.5136)

156. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 12 (Asia Cohort)
Description: Blood samples was collected for the assessment of hematology parameters. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 153
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 45 | 43 | 19 | 21
Grams per liter (g/L) | 2.3 (8.44) | 0.0 (8.45) | 1.4 (5.70) | -1.7 (7.31)

157. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Blood samples was collected for the assessment of hematology parameters. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 154
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Grams per liter (g/L)
  Week 24 | 3.2 (10.72) | -0.8 (9.81) | 2.4 (8.97)
  Week 52: number analyzed (Participants) | 29 | 28 | 15
  Week 52 | 1.9 (10.65) | -1.8 (9.95) | 2.4 (9.76)

158. Secondary Outcome: Change From Baseline in Hematology Parameter of Hemoglobin at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: Blood samples was collected for the assessment of hematology parameters. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Grams per liter (g/L)
  Week 24 | -0.5 (7.94) | -1.2 (8.77) | 3.3 (4.68)
  Week 52: number analyzed (Participants) | 4 | 5 | 6
  Week 52 | -0.5 (6.35) | -1.0 (11.51) | 2.5 (7.23)

159. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (AP), Gamma-Glutamyl Transpeptidase (GGT) at Week 12 (Asia Cohort)
Description: as for outcome 68
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 153
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 46 | 43 | 19 | 21
International units per liter (IU/L)
  Aspartate Aminotransferase | 3.5 (13.14) | 2.0 (5.29) | 2.9 (4.82) | 0.8 (8.26)
  Alanine Aminotransferase | 2.1 (16.90) | 2.5 (7.49) | 0.0 (7.85) | 2.8 (16.44)
  Alkaline Phosphatase | -1.9 (14.73) | -1.0 (11.52) | -4.2 (15.44) | -0.6 (16.52)
  Gamma-Glutamyl Transpeptidase | -3.0 (10.95) | 0.7 (12.28) | -3.5 (14.69) | 2.6 (12.52)

160. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of AST, ALT, AP, GGT at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 69
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 154
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
International units per liter (IU/L)
  AST. Week 24 | 0.1 (10.02) | 2.1 (6.20) | 3.2 (7.27)
  AST. Week 52: number analyzed (Participants) | 29 | 28 | 16
  AST. Week 52 | 0.9 (8.65) | 1.2 (5.34) | 4.2 (10.58)
  ALT, Week 24 | -1.0 (16.19) | 2.5 (8.56) | -0.2 (14.22)
  ALT, Week 52: number analyzed (Participants) | 29 | 28 | 16
  ALT, Week 52 | -2.3 (15.36) | -0.4 (5.95) | 2.0 (19.78)
  AP, Week 24 | -0.3 (15.15) | 0.3 (16.64) | -5.6 (15.14)
  AP, Week 52: number analyzed (Participants) | 29 | 28 | 16
  AP, Week 52 | -5.7 (15.00) | -6.3 (18.37) | -5.1 (21.76)
  GGT, Week 24 | -4.4 (9.83) | 0.7 (16.68) | -5.0 (17.60)
  GGT, Week 52: number analyzed (Participants) | 29 | 28 | 16
  GGT, Week 52 | -6.8 (10.38) | -2.1 (12.53) | 1.4 (20.96)

161. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of AST, ALT, AP, GGT at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 70
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
International units per liter (IU/L)
  AST, Week 24 | -0.5 (2.43) | -4.0 (9.14) | 4.3 (4.07)
  AST, Week 52: number analyzed (Participants) | 4 | 5 | 5
  AST, Week 52 | 1.3 (2.36) | -1.2 (1.64) | 2.6 (5.41)
  ALT, Week 24 | 0.5 (2.43) | -14.0 (25.91) | 1.7 (7.36)
  ALT, Week 52: number analyzed (Participants) | 4 | 5 | 5
  ALT, Week 52 | 6.0 (6.98) | -4.0 (5.92) | -2.0 (8.75)
  AP, Week 24 | -0.3 (7.74) | -6.0 (12.57) | 0.0 (26.44)
  AP, Week 52: number analyzed (Participants) | 4 | 5 | 5
  AP, Week 52 | -10.5 (18.16) | 1.6 (4.98) | -13.6 (21.48)
  GGT, Week 24 | -1.3 (5.75) | -10.8 (23.23) | -6.0 (12.94)
  GGT, Week 52: number analyzed (Participants) | 4 | 5 | 5
  GGT, Week 52 | 3.0 (6.78) | -4.0 (12.53) | -7.6 (15.45)

162. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 12 (Asia Cohort)
Description: as for outcome 71
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 153
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 46 | 43 | 19 | 21
Micromoles per liter (umol/L) | 0.2 (2.32) | 0.1 (2.64) | 1.1 (4.71) | -0.1 (2.68)

163. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 72
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: as for outcome 154
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Micromoles per liter (umol/L)
  Week 24 | 0.3 (2.60) | 0.2 (2.82) | 0.3 (3.79)
  Week 52: number analyzed (Participants) | 29 | 28 | 16
  Week 52 | 0.7 (2.69) | 1.6 (4.75) | 1.6 (2.85)

164. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Total Bilirubin at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 73
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Micromoles per liter (umol/L)
  Week 24 | -0.7 (1.97) | 3.2 (3.54) | 0.3 (2.75)
  Week 52: number analyzed (Participants) | 4 | 5 | 5
  Week 52 | 0.0 (1.41) | 2.0 (2.00) | 0.0 (1.41)

165. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 12 (Asia Cohort)
Description: Blood samples was collected for the assessment of clinical chemistry parameter albumin. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For the purpose of all analyses up to week 12, the placebo arms were pooled into a single placebo arm to primarily serve as a reference for the comparison of active treatment arms.
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 153
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 46 | 43 | 19 | 21
Grams per liter (g/L) | 0.8 (2.99) | -0.2 (2.26) | 2.1 (2.51) | -0.5 (2.68)

166. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 24 and Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: Blood samples was collected for the assessment of clinical chemistry parameter albumin. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value.
Time Frame: Baseline (Day 1), Week 24 and Week 52
Population: The analysis was performed on Safety Set participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 38 | 43 | 17
Grams per liter (g/L)
  Week 24 | 0.7 (2.81) | 0.3 (2.90) | 1.4 (4.01)
  Week 52: number analyzed (Participants) | 29 | 28 | 16
  Week 52 | 1.0 (2.54) | 0.2 (2.47) | 2.6 (3.50)

167. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter of Albumin at Week 24 and Week 52 for Placebo Switched Arms (Asia Cohort)
Description: Blood samples was collected for the assessment of clinical chemistry parameter albumin. Baseline was defined as latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting post dose visit value from Baseline value. For safety assessments baseline is interpreted as Week 12.
Time Frame: Baseline (Week 12), Week 24 and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 6 | 7
Grams per liter (g/L)
  Week 24 | 0.3 (3.01) | 1.2 (1.83) | 2.1 (2.54)
  Week 52: number analyzed (Participants) | 4 | 5 | 5
  Week 52 | 0.3 (1.71) | 2.0 (1.58) | 3.8 (3.70)

168. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 12 (Asia Cohort)
Description: as for outcome 77
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 77
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0

169. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 24 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 78
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 78
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0

170. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 24 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 79
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 78
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0

171. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 78
Time Frame: Baseline (Day 1) and Week 52
Population: The analysis was performed on the Safety Set participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 29 | 29 | 16
Millimoles per liter (mmol/L) | -0.166 (0.8128) | 0.146 (0.5227) | 0.743 (0.7569)

172. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Total Cholesterol at Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 81
Time Frame: Baseline (Week 4) and Week 52
Population: The analysis was performed on Safety Set-Placebo switch. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 4 | 5 | 5
Millimoles per liter (mmol/L) | 0.085 (0.4905) | 0.318 (1.4969) | 0.816 (0.5924)

173. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Low-density Lipoprotein (LDL) Cholesterol, High-density Lipoprotein (HDL) Cholesterol at Week 12 (Asia Cohort)
Description: as for outcome 82
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 77
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0

174. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 24 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 83
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 78
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0

175. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 24 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 84
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 78
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0

176. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 83
Time Frame: Baseline (Day 1) and Week 52
Population: as for outcome 171
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 29 | 29 | 16
Millimoles per liter (mmol/L)
  LDL cholesterol: number analyzed (Participants) | 28 | 29 | 16
  LDL cholesterol | -0.258 (0.7697) | 0.076 (0.4614) | 0.334 (0.4170)
  HDL cholesterol | -0.044 (0.2490) | -0.012 (0.2779) | 0.146 (0.3082)

177. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of LDL Cholesterol, HDL Cholesterol at Week 52 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 86
Time Frame: Baseline (Week 4) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 4 | 5 | 5
Millimoles per liter (mmol/L)
  LDL cholesterol | 0.218 (0.5604) | 0.094 (1.2936) | 0.438 (0.4544)
  HDL cholesterol | 0.000 (0.1089) | 0.042 (0.2400) | 0.226 (0.2204)

178. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 12 (Asia Cohort)
Description: as for outcome 87
Time Frame: Baseline (Day 1) and Week 12
Population: as for outcome 77
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0 | 0

179. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 24 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 88
Time Frame: Baseline (Day 1) and Week 24
Population: as for outcome 78
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0

180. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 24 for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 89
Time Frame: Baseline (Week 12) and Week 24
Population: as for outcome 78
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 0 | 0 | 0

181. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 52 for Treatment Arms Who Started Study Intervention From Day 1 (Asia Cohort)
Description: as for outcome 88
Time Frame: Baseline (Day 1) and Week 52
Population: The analysis was performed on the Safety Set participants who received study intervention from Day 01 to Week 52. Only those participants with data available at the indicated timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 29 | 29 | 16
Millimoles per liter (mmol/L) | 0.443 (1.4807) | 0.180 (0.4439) | 0.345 (0.6262)

182. Secondary Outcome: Change From Baseline in Lipid Profile Parameter of Triglycerides at Week 52 for Placebo Switched Arms (Asia Cohort)
Description: Blood samples was collected for the assessment of change from baseline in fasting lipid profile triglycerides levels. Baseline was defined as the latest pre-dose assessment with a non-missing value, including those from unscheduled visits. Change from Baseline was calculated by subtracting the post dose visit value from the Baseline value. For lipid profile assessments, baseline is interpreted as Week 4.
Time Frame: Baseline (Week 4) and Week 52
Population: as for outcome 64
Measure: Mean (Standard Deviation); unit: Millimoles per liter (mmol/L)
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 4 | 5 | 5
Millimoles per liter (mmol/L) | -0.288 (0.7348) | 0.398 (0.6266) | 0.328 (0.5965)

183. Secondary Outcome: Number of Participants With National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE)>=Grade 3 Hematological/Clinical Chemistry Abnormalities (Asia Cohort)
Description: Number of participants with NCI-CTCAE >=Grade 3 hematological/clinical chemistry abnormalities were summarized. Hematological and Clinical chemistry parameters were summarized according to the NCI-CTCAE, version 5.0: Grade 1: mild; Grade 2: moderate; Grade 3: severe; Grade 4: life-threatening or disabling. Higher grade indicates more severity. Data is presented for only those parameters for which participants had worst case >=Grade 3 shifts from Baseline.
Time Frame: Up to Week 59
Population: as for outcome 61
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asian Cohort)
Number analyzed (Participants) | 47 | 49 | 19 | 23
Participants
  Cholesterol - high, Total, Grade 3 | 1 | 0 | 0 | 0
  Lymphocyte count decreased, Total, Grade 3 | 1 | 1 | 2 | 0
  Hypertriglyceridemia, Total, Grade 3 | 1 | 1 | 1 | 0

184. Secondary Outcome: Concentrations of Granulocyte-macrophage Colony Stimulating Factor (GM-CSF) Autoantibody (Asia Cohort)
Description: as for outcome 93
Time Frame: At baseline
Population: The analysis was performed on the Safety Set. Only those participants with data available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: Microgram per liter (ug/L)
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0
Microgram per liter (ug/L) | 526.0 (NA) — NA indicate that data is not available since only one participant was analyzed, therefore Standard Deviation was not derived. |  |  |  |  |

185. Secondary Outcome: Number of Participants With Anti-GSK3196165 Antibodies (Asia Cohort)
Description: as for outcome 94
Time Frame: Up to Week 59
Population: The analysis was performed on the pharmacokinetic population which included participants in the Safety population who had at least 1 non-missing pharmacokinetic assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 47 | 49 | 19 | 6 | 8 | 9
Participants | 0 | 0 | 0 | 0 | 0 | 0

186. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) for Placebo Switched Arms (Global Cohort)
Description: as for outcome 152
Time Frame: Week 12 to Week 59
Population: The analysis was performed on Safety Set-Placebo switch for Placebo + MTX and GSK3196165 90 mg + MTX, Placebo + MTX and GSK3196165 150 mg + MTX, Placebo + MTX and Tofacitinib 5 mg + MTX (collected data from Week 12 to 59).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 85 | 80 | 67
Participants
  Participants with AE | 54 | 52 | 45
  Participants with SAE | 5 | 3 | 2
  Participants with AESI | 6 | 12 | 3

187. Secondary Outcome: Number of Participants With National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE)>=Grade 3 Hematological/Clinical Chemistry Abnormalities for Placebo Switched Arms (Global Cohort)
Description: as for outcome 183
Time Frame: Week 12 to Week 59
Population: as for outcome 186
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort)
Number analyzed (Participants) | 85 | 80 | 67
Participants
  Anemia, Total, Grade 3 | 0 | 2 | 1
  Lymphocyte count decreased, Grade 3 | 1 | 0 | 2
  Neutrophil count decreased, Total, Grade 3 | 0 | 1 | 0
  Lymphocyte count decreased, Grade 4 | 0 | 0 | 1
  Hypertriglyceridemia, Total, Grade 3 | 0 | 1 | 0

188. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESI) for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 152
Time Frame: Week 12 to Week 59
Population: as for outcome 186
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 8 | 8
Participants
  Participants with AE | 6 | 5 | 7
  Participants with SAE | 0 | 1 | 0
  Participants with AESI | 0 | 0 | 0

189. Secondary Outcome: Number of Participants With National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE)>=Grade 3 Hematological/Clinical Chemistry Abnormalities for Placebo Switched Arms (Asia Cohort)
Description: as for outcome 183
Time Frame: Week 12 to Week 59
Population: as for outcome 186
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
Number analyzed (Participants) | 6 | 8 | 8
Participants
  Cholesterol - high, Total, Grade 3 | 0 | 0 | 0
  Lymphocyte count decreased, Total, Grade 3 | 0 | 0 | 0
  Hypertriglyceridemia, Total, Grade 3 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: For both Global and Asian cohorts, AEs and SAEs were collected from the start of study intervention. For both cohorts, Pooled Placebo collected during the timeframe Week 0 to Week 12; Placebo+csDMARD and GSK3196165 90mg+csDMARD, Placebo+csDMARD and GSK3196165 150mg+csDMARD, Placebo+csDMARD and Tofacitinib 5mg+csDMARD collected during the timeframe Week 12 to Week 59; and GSK3196165 90mg+csDMARD, GSK3196165 150mg+csDMARD, Tofacitinib 5mg+csDMARD collected during the timeframe Week 0 to Week 59.
Description: The analysis was performed on the Safety Set for Pooled Placebo, GSK3196165 90 mg + MTX, GSK3196165 150 mg + MTX, Tofacitinib 5 mg + MTX. The analysis was performed on Safety Set-Period 2 for Placebo + MTX and GSK3196165 90 mg + MTX, Placebo + MTX and GSK3196165 150 mg + MTX, Placebo + MTX and Tofacitinib 5 mg + MTX.
Arm/Group | GSK3196165 90mg + csDMARD (Global Cohort) | GSK3196165 150mg + csDMARD (Global Cohort) | Tofacitinib 5mg + csDMARD (Global Cohort) | Pooled Placebo (Global Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort) | GSK3196165 90mg + csDMARD (Asia Cohort) | GSK3196165 150mg + csDMARD (Asia Cohort) | Tofacitinib 5mg + csDMARD (Asia Cohort) | Pooled Placebo (Asia Cohort) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort)
All-Cause Mortality (participants affected / at risk) | 5/545 | 6/539 | 2/286 | 0/255 | 1/85 | 1/80 | 0/67 | 0/47 | 0/49 | 0/19 | 0/23 | 0/6 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 44/545 | 43/539 | 31/286 | 6/255 | 5/85 | 3/80 | 2/67 | 5/47 | 4/49 | 2/19 | 1/23 | 0/6 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 233/545 | 208/539 | 105/286 | 3/255 | 28/85 | 31/80 | 23/67 | 28/47 | 39/49 | 18/19 | 10/23 | 6/6 | 5/8 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3196165 90mg + csDMARD (Global Cohort) (N=545) | GSK3196165 150mg + csDMARD (Global Cohort) (N=539) | Tofacitinib 5mg + csDMARD (Global Cohort) (N=286) | Pooled Placebo (Global Cohort) (N=255) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) (N=85) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) (N=80) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort) (N=67) | GSK3196165 90mg + csDMARD (Asia Cohort) (N=47) | GSK3196165 150mg + csDMARD (Asia Cohort) (N=49) | Tofacitinib 5mg + csDMARD (Asia Cohort) (N=19) | Pooled Placebo (Asia Cohort) (N=23) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) (N=6) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) (N=8) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort) (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus node dysfunction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ulcerative keratitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mesenteric cyst (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Secondary amyloidosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 5 (5) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia cryptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint destruction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colorectal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
IgA nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrosalpinx (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cervix carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK3196165 90mg + csDMARD (Global Cohort) (N=545) | GSK3196165 150mg + csDMARD (Global Cohort) (N=539) | Tofacitinib 5mg + csDMARD (Global Cohort) (N=286) | Pooled Placebo (Global Cohort) (N=255) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Global Cohort) (N=85) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Global Cohort) (N=80) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Global Cohort) (N=67) | GSK3196165 90mg + csDMARD (Asia Cohort) (N=47) | GSK3196165 150mg + csDMARD (Asia Cohort) (N=49) | Tofacitinib 5mg + csDMARD (Asia Cohort) (N=19) | Pooled Placebo (Asia Cohort) (N=23) | Placebo + csDMARD and GSK3196165 90mg + csDMARD (Asia Cohort) (N=6) | Placebo + csDMARD and GSK3196165 150mg + csDMARD (Asia Cohort) (N=8) | Placebo + csDMARD and Tofacitinib 5mg + csDMARD (Asia Cohort) (N=8)
Anaemia (Blood and lymphatic system disorders) | 35 (41) | 19 (20) | 8 (9) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 4 (4) | 7 (8) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 33 (45) | 38 (57) | 24 (32) | 0 (0) | 8 (9) | 3 (5) | 4 (5) | 0 (0) | 5 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scleritis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Salivary gland mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 42 (112) | 47 (137) | 5 (7) | 3 (3) | 5 (8) | 10 (15) | 0 (0) | 2 (5) | 5 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 49 (51) | 32 (35) | 27 (27) | 0 (0) | 3 (3) | 4 (4) | 8 (8) | 2 (2) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 28 (33) | 33 (43) | 15 (15) | 0 (0) | 5 (7) | 1 (1) | 5 (8) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 4 (5) | 1 (1) | 4 (4) | 7 (10) | 3 (8) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 34 (47) | 39 (45) | 19 (24) | 0 (0) | 2 (3) | 6 (6) | 1 (1) | 1 (1) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (10) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood beta-D-glucan increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Lipids abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (13) | 6 (9) | 1 (1) | 2 (3) | 0 (0) | 1 (4) | 3 (4)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (7) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (7) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 41 (51) | 40 (53) | 20 (23) | 0 (0) | 3 (4) | 5 (7) | 6 (7) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 33 (36) | 19 (23) | 13 (15) | 0 (0) | 4 (5) | 5 (6) | 5 (5) | 1 (3) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post herpetic neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 30 (32) | 31 (32) | 19 (20) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-01-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03970837/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT03970837/SAP_001.pdf